CLINICAL TRIAL: NCT01041404
Title: A Randomized, Open-label Study of the Effect of First-line Herceptin in Combination With a Fluoropyrimidine and Cisplatin Versus Chemotherapy Alone on Overall Survival in Patients With HER2-positive Advanced Gastric Cancer
Brief Title: ToGA Study - A Study of Herceptin (Trastuzumab) in Combination With Chemotherapy Compared With Chemotherapy Alone in Patients With HER2-Positive Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO18255
Record Dates: First submitted 2009-12-29; First posted 2009-12-31 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Fluorouracil; Cisplatin; Capecitabine

ARMS (2):
- Trastuzumab, Fluoropyrimidine, Cisplatin (Experimental): Participants received an initial loading dose of 8 milligrams per kilogram (mg/kg) trastuzumab i.v. on Day 1 of cycle, followed by 6 mg/kg i.v. every 3 weeks until disease progression; 800 mg/m2 fluorouracil i.v. on Days 1 through 5 of cycle every 3 weeks for 6 cycles; 80 mg/m2 cisplatin i.v. on Day 1 of cycle every 3 weeks for 6 cycles; and 1000 mg/m2 capecitabine p.o. twice daily on Days 1 through 15 of cycle every 3 weeks for 6 cycles.
  Interventions: Drug: Trastuzumab; Drug: Fluorouracil; Drug: Cisplatin; Drug: Capecitabine
- Fluoropyrimidine, Cisplatin (Active Comparator): Participants received 800 milligrams per square meter (mg/m2) fluorouracil intravenous (i.v.) on Days 1 through 5 of cycle every 3 weeks for 6 cycles; 80 mg/m2 cisplatin i.v. on Day 1 of cycle every 3 weeks for 6 cycles; and 1000 mg/m2 capecitabine orally (p.o.) twice daily on Days 1 through 15 of cycle every 3 weeks for 6 cycles.
  Interventions: Drug: Fluorouracil; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Trastuzumab — Initial loading dose 8 mg/kg i.v. infusion on Day 1 of cycle, followed by 6 mg/kg i.v. infusion every 3 weeks until disease progression
  Other Names: Herceptin
  Arms: Trastuzumab, Fluoropyrimidine, Cisplatin
Drug: Fluorouracil — 800 mg/m2 i.v. infusion on Days 1 through 5 of cycle every 3 weeks for 6 cycles
  Other Names: 5-FU
Drug: Cisplatin — 80 mg/m2 i.v. infusion on Day 1 of cycle every 3 weeks for 6 cycles
Drug: Capecitabine — 1000 mg/m2 p.o. twice daily on Days 1 through 15 of cycle every 3 weeks for 6 cycles
  Other Names: Xeloda

SUMMARY:
This parallel, randomized, open-label, multi-centre study will evaluate the effect on overall survival of trastuzumab (Herceptin) in combination with a chemotherapy compared to the chemotherapy alone in patients with HER2-positive advanced gastric cancer. Trastuzumab (Herceptin) will be administered as intravenous infusion of 6 mg/kg (loading dose 8 mg/kg) every 3 weeks. The chemotherapy consists of a combination of 6 cycles of fluorouracil (800 mg/m2/day intravenous infusion every 3 weeks) and cisplatin (80 mg/m2 intravenous infusion every 3 weeks), or capecitabine (Xeloda, 1000 mg/m2 po twice daily for 14 days every 3 weeks) and cisplatin (80 mg/m2 intravenous infusion every 3 weeks). Treatment with trastuzumab (Herceptin) will continue until disease progression. The target sample size is 300-600 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >=18 years of age
* Inoperable locally advanced, recurrent, and/or metastatic cancer of the stomach or gastro-esophageal junction
* Adenocarcinoma
* HER2-positive tumors

Exclusion Criteria:

* Previous chemotherapy for advanced/metastatic disease
* Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome
* History of cardiac disease
* Dyspnoea at rest, due to complications of advanced malignancy or other disease, or patients who require supportive oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (107):
- Australia (6):
  - Adelaide
  - Kurralta Park
  - Melbourne
  - Milton
  - Perth
  - Sydney
- Leuven, Belgium
- Brazil (3):
  - Barretos
  - Rio de Janeiro
  - São Paulo
- China (8):
  - Beijing
  - Guangdong
  - Guangzhou
  - Jiangsu
  - Nanjing
  - Shanghai
  - Suzhou
  - Wuhan
- San José, Costa Rica
- Denmark (2):
  - Herlev
  - Odense
- Tampere, Finland
- France (8):
  - Brest
  - Caen
  - Colmar
  - Lille
  - Marseille
  - Reims
  - Rouen
  - Strasbourg
- Germany (5):
  - Heidelberg
  - Mainz
  - München
  - Trier
  - Witten
- Guatemala City, Guatemala
- India (4):
  - Hyderabad
  - Kochi
  - Mumbai
  - New Delhi
- Italy (6):
  - Ancona
  - Florence
  - Napoli
  - Parma
  - Roma
  - Udine
- Japan (12):
  - Aichi
  - Chiba
  - Ehime
  - Fukuoka
  - Hyōgo
  - Nagano
  - Osaka
  - Saitama
  - Shizuoka
  - Tochigi
  - Tokyo
  - Yamagata
- Mexico (4):
  - Guadalajara
  - Mexico City
  - Mérida
  - Monterrey
- Panama City, Panama
- Peru (2):
  - Callao
  - Lima
- Portugal (6):
  - Braga
  - Coimbra
  - Faro
  - Guimarães
  - Lisbon
  - Porto
- Russia (10):
  - Chelyabinsk
  - Ivanovo
  - Kazan'
  - Moscow
  - Ryazan
  - Saint Petersburg
  - Samara
  - Ufa
  - Yaroslavl
  - Yekaterinburg
- South Africa (2):
  - Cape Town
  - Durban
- South Korea (6):
  - Buchun
  - Bundang City
  - Daegu
  - Goyang-si
  - Pusan
  - Seoul
- Spain (4):
  - Barcelona
  - Girona
  - Madrid
  - Valencia
- Taiwan (3):
  - Changhua
  - Kaohsiung City
  - Taipei
- Turkey (Türkiye) (3):
  - Istanbul
  - Izmir
  - Shhiye, Ankara
- United Kingdom (8):
  - Birmingham
  - Denbigh
  - Dundee
  - Glasgow
  - Manchester
  - Metropolitan Borough of Wirral
  - Weston-super-Mare
  - Wolverhampton

REFERENCES:
- [Derived] Van Cutsem E, Bang YJ, Feng-Yi F, Xu JM, Lee KW, Jiao SC, Chong JL, Lopez-Sanchez RI, Price T, Gladkov O, Stoss O, Hill J, Ng V, Lehle M, Thomas M, Kiermaier A, Ruschoff J. HER2 screening data from ToGA: targeting HER2 in gastric and gastroesophageal junction cancer. Gastric Cancer. 2015 Jul;18(3):476-84. doi: 10.1007/s10120-014-0402-y. Epub 2014 Jul 20. PMID 25038874
- [Derived] Satoh T, Bang YJ, Gotovkin EA, Hamamoto Y, Kang YK, Moiseyenko VM, Ohtsu A, Van Cutsem E, Al-Sakaff N, Urspruch A, Hill J, Weber HA, Chung HC; ToGA Trial Investigators. Quality of life in the trastuzumab for gastric cancer trial. Oncologist. 2014 Jul;19(7):712-9. doi: 10.1634/theoncologist.2014-0058. Epub 2014 Jun 20. PMID 24951609
- [Derived] Satoh T, Omuro Y, Sasaki Y, Hamamoto Y, Boku N, Tamura T, Ohtsu A. Pharmacokinetic analysis of capecitabine and cisplatin in combination with trastuzumab in Japanese patients with advanced HER2-positive gastric cancer. Cancer Chemother Pharmacol. 2012 Apr;69(4):949-55. doi: 10.1007/s00280-011-1783-9. Epub 2011 Nov 25. PMID 22116464
- [Derived] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoropyrimidine/Cisplatin (FP): Participants received fluoropyrimidine (EITHER 5-fluorouracil [5-FU] or capecitabine, at the investigator's discretion) and cisplatin once every 3 weeks (one cycle) for a maximum of 6 cycles as follows: cisplatin 80 milligrams per square meter (mg/m^2), intravenously (IV), on Day 1 and EITHER: 5-FU 800 mg/m^2 continuous IV infusion on Days 1 through 5 OR capecitabine 1000 mg/m^2 tablets, orally (PO), twice daily (BID) from the evening of Day 1 through the morning of Day 15.
- Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H): Participants received trastuzumab plus fluoropyrimidine (EITHER 5-FU or capecitabine, at the investigator's discretion) and cisplatin once every 3 weeks (one cycle) for a maximum of 6 cycles (except as noted) as follows: trastuzumab 8 milligrams per kilogram (mg/kg), IV, on Day 1 (Cycle 1), followed by 6 mg/kg, IV (Cycles 2 onward, administered until disease progression); cisplatin 80 mg/m^2 IV on Day 1; and EITHER 5-FU 800 mg/m^2 continuous IV infusion on Days 1 through 5 OR capecitabine 1000 mg/m^2 tablets, PO BID from the evening of Day 1 through the morning of Day 15.
Period: Overall Study
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Started | 290 | 294
Entered Follow-Up | 251 | 251
Died in Follow-up | 199 | 200
Lost to Follow-up | 12 | 10
Alive in Follow-up | 40 | 41
Completed | 0 (Summary of withdrawals represents withdrawals from treatment, rather than withdrawals from study.) | 0 (Summary of withdrawals represents withdrawals from treatment, rather than withdrawals from study.)
Not Completed | 290 | 294
Not completed — Adverse Event | 45 | 35
Not completed — Lack of Efficacy | 200 | 210
Not completed — Violation of Selection Criteria | 0 | 1
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 29 | 23
Not completed — Failure to Return | 1 | 2
Not completed — Other | 11 | 23

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Fluoropyrimidine/Cisplatin (FP): Participants received fluoropyrimidine (EITHER 5-FU or capecitabine, at the investigator's discretion) and cisplatin once every 3 weeks (one cycle) for a maximum of 6 cycles as follows: cisplatin 80 mg/m^2, IV, on Day 1 and EITHER: 5-FU 800 mg/m^2 continuous IV infusion on Days 1 through 5 OR capecitabine 1000 mg/m^2, tablets, PO, BID from the evening of Day 1 through the morning of Day 15.
- Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H): Participants received trastuzumab plus fluoropyrimidine (EITHER 5-FU or capecitabine, at the investigator's discretion) and cisplatin once every 3 weeks (one cycle) for a maximum of 6 cycles (except as noted) as follows: trastuzumab 8 mg/kg, IV, on Day 1 (Cycle 1), followed by 6 mg/kg, IV (Cycles 2 onward, administered until disease progression); cisplatin 80 mg/m^2 IV on Day 1; and EITHER 5-FU 800 mg/m^2 continuous IV infusion on Days 1 through 5 OR capecitabine 1000 mg/m^2 tablets, PO BID from the evening of Day 1 through the morning of Day 15.
- Total: Total of all reporting groups
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H) | Total
Number analyzed (Participants) | 290 | 294 | 584
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.22) | 59.4 (10.75) | 59.0 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 68 | 140
  Male | 218 | 226 | 444

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Participants were censored at the last date of tumor measurement, the last date in the study drug log, or the date of last follow-up.
Time Frame: Baseline (BL), Days 1, 8, 15, 22, 43, 64, 85, 106, 127, and every 21 days until the end of study, 1 year after the cut-off date for the 2nd interim efficacy analysis
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
percentage of participants | 62.8 | 56.8

2. Secondary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of progressive disease (PD) or date of death, whichever occurs first. For target lesions (TL), PD was defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD) of TLs, taking as a reference the smallest SLD recorded since the treatment started, or the appearance of one or more lesions. For non-target lesions (NTL), PD was defined as an unequivocal progression of existing NTLs. Participants were censored at the last date of tumor measurement, the last date in the study drug log, or the date of last follow-up.
Time Frame: BL, Days 43, 85, and 127, and every 21 days thereafter until disease progression or the end of study, 1 year after the cut-off date for the 2nd interim efficacy analysis
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
percentage of participants | 81.0 | 76.9

3. Secondary Outcome: Progression-Free Survival - Time to Event
Description: The median time, in months, from the date of randomization to the date of a PFS event. Participants were censored at the last date of tumor measurement, the last date in the study drug log, or the date of last follow-up.
Time Frame: as for outcome 2
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Fluoropyrimidine, Cisplatin: Participants received fluorouracil 800 mg/m^2 IV on Days 1 through 5 of cycle every 3 weeks for 6 cycles. Participants also received cisplatin 80 mg/m^2, IV, on Day 1 of cycle every 3 weeks for 6 cycles; as well as, capecitabine 1000 mg/m^2, PO, twice daily on Days 1 through 15 of cycle every 3 weeks for 6 cycles.
- Trastuzumab, Fluoropyrimidine, Cisplatin: Participants received an initial loading dose of trastuzumab 8 mg/kg, IV, on Day 1 of cycle, followed by 6 mg/kg, IV, every 3 weeks until disease progression. Participants also received fluorouracil 800 mg/m^2 IV on Days 1 through 5 of cycle every 3 weeks for 6 cycles; cisplatin 80 mg/m^2 IV on Day 1 of cycle every 3 weeks for 6 cycles; and capecitabine 1000 mg/m^2 PO twice daily on Days 1 through 15 of cycle every 3 weeks for 6 cycles.
Arm/Group | Fluoropyrimidine, Cisplatin | Trastuzumab, Fluoropyrimidine, Cisplatin
Number analyzed (Participants) | 290 | 294
months | 5.5 [5 to 6] | 6.7 [6 to 8]
Statistical Analysis 1: Comparison: Fluoropyrimidine, Cisplatin vs Trastuzumab, Fluoropyrimidine, Cisplatin; Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.59 to 0.85]

4. Secondary Outcome: Time to Progression (TTP) - Percentage of Participants With an Event
Description: TTP was defined as the time from the date of randomization and the date of the first occurrence of PD. Participants were censored at the last date of tumor assessment, the last date in the study drug log, or the last date of follow-up.
Time Frame: as for outcome 2
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
percentage of participants | 74.1 | 70.7

5. Secondary Outcome: Time to Progression - Time to Event
Description: The median time, in months, from the date of randomized to the date of a TTP event. Participants were censored at the last date of tumor assessment, the last date in the study drug log, or the last date of follow-up.
Time Frame: as for outcome 2
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
months | 5.6 [5 to 6] | 7.1 [6 to 8]
Statistical Analysis 1: Comparison: Fluoropyrimidine/Cisplatin (FP) vs Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H); Test type: Superiority or Other; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.58 to 0.85]

6. Secondary Outcome: Percentage of Participants With Confirmed Complete Response (CR) or Partial Response (PR) Determined by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: For TLs, a CR was defined as the disappearance of all TLs and a PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline SLD. For NTLs, a CR was defined as the disappearance of all NTLs and normalization of tumor marker levels.
Time Frame: as for outcome 2
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
percentage of participants | 34.5 [29.0 to 40.3] | 47.3 [41.5 to 53.2]
Statistical Analysis 1: Comparison: Fluoropyrimidine/Cisplatin (FP) vs Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H); Test type: Superiority or Other; p = 0.0017, Chi-squared; Difference in Response Rates = 12.80, 95% CI 2-sided [4.7 to 20.9]

7. Secondary Outcome: Duration of Response - Percentage of Participants With an Event
Description: Duration of response was defined for responders as the time from the date on which the CR or PR was first recorded to the date on which PD is first noted. Participants were censored on the date of death, the date of last tumor measurement, the last date in study drug log, or the date of last follow-up.
Time Frame: as for outcome 2
Population: FAS; only participants with a CR or PR were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 100 | 139
percentage of participants | 80.0 | 71.9

8. Secondary Outcome: Duration of Response
Description: The median time, in months, of the duration of response. Participants were censored at the date of death, the date of last tumor measurement, the last date in study drug log, or the date of last follow-up.
Time Frame: as for outcome 2
Population: FAS; only participants with a CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 100 | 139
months | 4.8 [4 to 6] | 6.9 [6 to 8]
Statistical Analysis 1: Comparison: Fluoropyrimidine/Cisplatin (FP) vs Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H); Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.40 to 0.73]

9. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit was defined as stable disease (SD), CR, or PR for 6 weeks or longer as determined by RECIST. For TLs, SD was defined as neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD, taking as a reference the smallest SLD recorded since treatment had started. For NTLs, SD was defined as a persistence of one or more NTLs and/or maintenance of tumor marker levels above the normal limits.
Time Frame: as for outcome 2
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
percentage of participants | 69.3 [63.7 to 74.6] | 78.9 [73.8 to 83.4]
Statistical Analysis 1: Comparison: Fluoropyrimidine/Cisplatin (FP) vs Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H); Test type: Superiority or Other; p = 0.0081, Chi-squared; Difference in Clinical Benefit Rate = 9.60, 95% CI 2-sided [2.4 to 16.9]
Statistical Analysis 2: Comparison: Fluoropyrimidine/Cisplatin (FP) vs Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H); Test type: Superiority or Other; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.14 to 2.41]

10. Primary Outcome: Overall Survival - Time to Event
Description: The median time, in months, from the date of randomization to the date of an OS event. Participants were censored at the last date tumor measurement, the last date in the study drug log, or the date of last follow-up.
Time Frame: BL, Days 1, 8, 15, 22, 43, 64, 85, 106, 127, and every 21 days until the end of study, 1 year after the cut-off date for the 2nd interim efficacy analysis
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
months | 11.1 [10 to 13] | 13.8 [12 to 16]
Statistical Analysis 1: Comparison: Fluoropyrimidine/Cisplatin (FP) vs Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H); Test type: Superiority or Other; p = 0.0046, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.60 to 0.91]

11. Secondary Outcome: European Organisation For the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ C-30) Questionnaire Scores
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score equals (=) better level of functioning or greater degree of symptoms.
Time Frame: BL, Days 1, 22, 43, 64, 85, 106, 127, and every 21 days until disease progression of the end of study, 1 year after the cut-off date for the 2nd interim efficacy analysis
Population: FAS; n (number) = number of participants assessed for a specific parameter at a given visit.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
scores on a scale
  Global Health Status: BL (n=274,287) | 55.3 (1.43) | 54.9 (1.30)
  Global Health Status: Week 4 (n=235,249) | 61.0 (1.37) | 60.9 (1.28)
  Global Health Status: Week 7 (n=180,220) | 60.9 (1.54) | 60.5 (1.36)
  Global Health Status: Week 10 (n=176,202) | 62.3 (1.58) | 61.9 (1.42)
  Global Health Status: Week 13 (n=152,182) | 63.8 (1.77) | 63.6 (1.47)
  Global Health Status: Week 16 (n=121,165) | 60.8 (1.85) | 61.9 (1.58)
  Global Health Status: Week 19 (n=114,143) | 61.0 (1.94) | 63.8 (1.80)
  Global Health Status: Week 22 (n=78,143) | 65.1 (2.32) | 64.9 (1.76)
  Global Health Status: Week 25 (n=64,124) | 68.0 (2.65) | 67.8 (2.02)
  Global Health Status: Week 28 (n=47,111) | 72.0 (2.69) | 68.5 (2.08)
  Global Health Status: Week 31 (n=45,95) | 69.6 (2.83) | 70.0 (2.07)
  Global Health Status: Week 34 (n=36,87) | 70.8 (3.55) | 72.0 (2.18)
  Global Health Status: Week 37 (n=29,64) | 66.1 (3.72) | 70.6 (2.41)
  Global Health Status: Week 40 (n=23,55) | 62.0 (4.97) | 70.6 (2.92)
  Global Health Status: Week 43 (n=12,43) | 72.9 (5.14) | 73.6 (3.23)
  Global Health Status: Week 46 (n=13,42) | 75.0 (4.00) | 73.8 (3.18)
  Global Health Status: Week 49 (n=9,36) | 68.5 (5.69) | 76.6 (2.83)
  Global Health Status: Week 52 (n=7,29) | 72.6 (3.95) | 71.3 (4.02)
  Global Health Status: Week 55 (n=5,24) | 76.7 (4.08) | 73.8 (4.68)
  Global Health Status: Week 58 (n=5,21) | 76.7 (4.08) | 73.8 (4.68)
  Global Health Status: Week 61 (n=4,17) | 79.2 (7.98) | 72.5 (5.48)
  Global Health Status: Week 64 (n=3,20) | 77.8 (5.56) | 70.0 (4.85)
  Global Health Status: Week 67 (n=4,17) | 75.0 (4.81) | 72.5 (5.14)
  Global Health Status: Week 70 (n=3,14) | 77.8 (5.56) | 68.5 (5.61)
  Global Health Status: Week 73 (n=3,12) | 80.6 (2.78) | 68.1 (5.97)
  Global Health Status: Week 76 (n=3,8) | 77.8 (5.56) | 67.7 (8.97)
  Global Health Status: Week 79 (n=3,9) | 77.8 (5.56) | 69.4 (7.08)
  Global Health Status: Week 82 (n=2,5) | 83.3 (0.00) | 60.0 (10.34)
  Global Health Status: Week 85 (n=2,6) | 83.3 (0.00) | 79.2 (6.72)
  Global Health Status: Week 88 (n=2,6) | 83.3 (0.00) | 73.6 (5.45)
  Global Health Status: Week 91 (n=2,4) | 83.3 (0.00) | 79.2 (5.38)
  Global Health Status: Week 94 (n=2,6) | 83.3 (0.00) | 79.2 (7.98)
  Global Health Status: Week 97 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 78.3 (3.33)
  Global Health Status: Week 100 (n=1,4) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 85.4 (5.24)
  Global Health Status: Week 103 (n=1,3) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 75.0 (4.81)
  Global Health Status: Week 106 (n=1,4) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 77.1 (3.99)
  Global Health Status: Week 109 (n=1,4) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 77.1 (3.99)
  Global Health Status: Week 112 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 75.0 (3.73)
  Global Health Status: Week 115 (n=1,4) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 72.9 (3.99)
  Global Health Status: Week 118 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 75.0 (3.73)
  Global Health Status: Week 121 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 75.0 (3.73)
  Global Health Status: Week 124 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 81.7 (5.53)
  Global Health Status: Week 127 (n=1,3) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 72.2 (5.56)
  Global Health Status: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 72.2 (5.56)
  Global Health Status: Week 133 (n=1,3) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 72.2 (5.56)
  Global Health Status: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 66.7 (0.00)
  Global Health Status: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 66.7 (0.00)
  Global Health Status: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 66.7 (0.00)
  Global Health Status: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 66.7 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Global Health Status: Final Visit (n=158,160) | 53.2 (2.09) | 53.1 (2.20)
  Physical Functioning: BL (n=276,287) | 78.9 (1.16) | 79.6 (1.17)
  Physical Functioning: Week 4 (n=235,250) | 76.0 (1.27) | 79.5 (1.20)
  Physical Functioning: Week 7 (n=181,220) | 79.3 (1.37) | 79.3 (1.25)
  Physical Functioning: Week 10 (n=174,201) | 78.2 (1.47) | 80.2 (1.22)
  Physical Functioning: Week 13 (n=151,183) | 80.2 (1.53) | 80.5 (1.36)
  Physical Functioning: Week 16 (n=121,165) | 79.8 (1.58) | 80.7 (1.37)
  Physical Functioning: Week 19 (n=114,143) | 78.8 (1.81) | 81.5 (1.49)
  Physical Functioning: Week 22 (n=79,143) | 80.7 (2.20) | 83.6 (1.38)
  Physical Functioning: Week 25 (n=64,124) | 85.8 (2.07) | 84.8 (1.30)
  Physical Functioning: Week 28 (n=47,110) | 86.2 (2.50) | 83.7 (1.60)
  Physical Functioning: Week 31 (n=45,95) | 85.6 (2.45) | 85.4 (1.66)
  Physical Functioning: Week 34 (n=37,87) | 86.3 (2.50) | 85.1 (1.89)
  Physical Functioning: Week 37 (n=29,64) | 85.7 (3.43) | 85.8 (2.05)
  Physical Functioning: Week 40 (n=24,55) | 84.4 (3.51) | 88.2 (1.88)
  Physical Functioning: Week 43 (n=12,43) | 85.6 (3.75) | 89.9 (1.85)
  Physical Functioning: Week 46 (n=14,42) | 87.6 (3.03) | 91.9 (1.53)
  Physical Functioning: Week 49 (n=10,36) | 88.7 (3.45) | 92.0 (1.61)
  Physical Functioning: Week 52 (n=8,30) | 88.3 (3.93) | 89.2 (2.71)
  Physical Functioning: Week 55 (n=6,24) | 85.6 (5.28) | 93.1 (1.90)
  Physical Functioning: Week 58 (n=6,21) | 86.7 (5.71) | 91.4 (2.88)
  Physical Functioning: Week 61 (n=4,17) | 91.7 (5.00) | 91.0 (3.66)
  Physical Functioning: Week 64 (n=3,20) | 95.6 (4.44) | 91.0 (3.36)
  Physical Functioning: Week 67 (n=4,17) | 93.3 (4.71) | 93.3 (2.56)
  Physical Functioning: Week 70 (n=3,14) | 97.8 (2.22) | 92.9 (3.73)
  Physical Functioning: Week 73 (n=3,12) | 97.8 (2.22) | 91.1 (3.70)
  Physical Functioning: Week 76 (n=3,8) | 95.6 (4.44) | 90.0 (5.49)
  Physical Functioning: Week 79 (n=3,9) | 95.6 (4.44) | 92.6 (3.41)
  Physical Functioning: Week 82 (n=2,6) | 93.3 (6.67) | 90.0 (6.38)
  Physical Functioning: Week 85 (n=2,6) | 100.0 (0.00) | 95.6 (2.81)
  Physical Functioning: Week 88 (n=2,6) | 100.0 (0.00) | 95.6 (2.22)
  Physical Functioning: Week 91 (n=2,4) | 100.0 (0.00) | 98.3 (1.67)
  Physical Functioning: Week 94 (n=2,6) | 100.0 (0.00) | 97.8 (2.22)
  Physical Functioning: Week 97 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 97.3 (2.67)
  Physical Functioning: Week 100 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.7 (3.33)
  Physical Functioning: Week 103 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.7 (3.33)
  Physical Functioning: Week 106 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 98.3 (1.67)
  Physical Functioning: Week 109 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.0 (3.19)
  Physical Functioning: Week 112 (n=1,5) | 93.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 97.3 (2.67)
  Physical Functioning: Week 115 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 93.3 (4.71)
  Physical Functioning: Week 118 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.0 (4.00)
  Physical Functioning: Week 121 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 94.7 (3.89)
  Physical Functioning: Week 124 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.0 (2.67)
  Physical Functioning: Week 127 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 93.3 (3.85)
  Physical Functioning: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 93.3 (6.67)
  Physical Functioning: Week 133 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.6 (4.44)
  Physical Functioning: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 93.3 (6.67)
  Physical Functioning: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 93.3 (6.67)
  Physical Functioning: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 93.3 (6.67)
  Physical Functioning: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Physical Functioning: Final Visit (n=158,161) | 72.1 (1.97) | 73.8 (2.19)
  Role Functioning: BL (n=276,287) | 73.2 (1.70) | 73.9 (1.68)
  Role Functioning: Week 4 (n=234,250) | 67.4 (1.85) | 76.1 (1.67)
  Role Functioning: Week 7 (n=181,220) | 70.9 (1.99) | 73.3 (1.85)
  Role Functioning: Week 10 (n=176,202) | 70.2 (2.06) | 74.3 (1.87)
  Role Functioning: Week 13 (n=152,182) | 73.4 (2.11) | 75.1 (1.93)
  Role Functioning: Week 16 (n=121,165) | 72.0 (2.41) | 74.6 (1.98)
  Role Functioning: Week 19 (n=114,143) | 71.1 (2.21) | 75.8 (2.10)
  Role Functioning: Week 22 (n=79,142) | 74.7 (2.81) | 79.7 (1.93)
  Role Functioning: Week 25 (n=64,124) | 81.3 (2.93) | 82.4 (1.99)
  Role Functioning: Week 28 (n=47,110) | 80.5 (3.52) | 79.7 (2.17)
  Role Functioning: Week 31 (n=45,95) | 82.2 (2.87) | 81.1 (2.45)
  Role Functioning: Week 34 (n=37,87) | 83.3 (3.10) | 82.2 (2.64)
  Role Functioning: Week 37 (n=29,64) | 81.6 (4.16) | 81.5 (2.90)
  Role Functioning: Week 40 (n=24,55) | 79.9 (4.91) | 82.1 (3.11)
  Role Functioning: Week 43 (n=12,43) | 80.6 (4.95) | 86.8 (2.63)
  Role Functioning: Week 46 (n=14,42) | 82.1 (4.44) | 86.5 (2.74)
  Role Functioning: Week 49 (n=10,36) | 81.7 (6.78) | 88.0 (2.94)
  Role Functioning: Week 52 (n=8,30) | 85.4 (5.84) | 84.4 (3.57)
  Role Functioning: Week 55 (n=6,24) | 80.6 (5.12) | 88.2 (3.68)
  Role Functioning: Week 58 (n=6,21) | 77.8 (5.56) | 89.7 (3.14)
  Role Functioning: Week 61 (n=4,17) | 83.3 (9.62) | 87.3 (4.17)
  Role Functioning: Week 64 (n=3,20) | 83.3 (9.62) | 87.5 (4.17)
  Role Functioning: Week 67 (n=4,17) | 83.3 (6.80) | 90.2 (3.52)
  Role Functioning: Week 70 (n=3,14) | 88.9 (5.56) | 86.9 (5.00)
  Role Functioning: Week 73 (n=3,12) | 88.9 (5.56) | 80.6 (5.36)
  Role Functioning: Week 76 (n=3,8) | 83.3 (9.62) | 81.3 (7.34)
  Role Functioning: Week 79 (n=3,9) | 83.3 (9.62) | 81.5 (7.58)
  Role Functioning: Week 82 (n=2,6) | 91.7 (8.33) | 80.6 (10.90)
  Role Functioning: Week 85 (n=2,6) | 100.0 (0.00) | 91.7 (5.69)
  Role Functioning: Week 88 (n=2,6) | 91.7 (8.33) | 94.4 (5.56)
  Role Functioning: Week 91 (n=2,4) | 91.7 (8.33) | 91.7 (8.33)
  Role Functioning: Week 94 (n=2,6) | 100.0 (0.00) | 100.0 (0.00)
  Role Functioning: Week 97 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 90.0 (6.67)
  Role Functioning: Week 100 (n=1,4) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 100.0 (0.00)
  Role Functioning: Week 103 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 100.0 (0.00)
  Role Functioning: Week 106 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 100.0 (0.00)
  Role Functioning: Week 109 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.8 (4.17)
  Role Functioning: Week 112 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 93.3 (6.67)
  Role Functioning: Week 115 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 83.3 (9.62)
  Role Functioning: Week 118 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 86.7 (8.16)
  Role Functioning: Week 121 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 90.0 (6.67)
  Role Functioning: Week 124 (n=1,5) | 83.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 90.0 (6.67)
  Role Functioning: Week 127 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 88.9 (11.11)
  Role Functioning: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 88.9 (11.11)
  Role Functioning: Week 133 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 88.9 (11.11)
  Role Functioning: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 83.3 (16.67)
  Role Functioning: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 83.3 (16.67)
  Role Functioning: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 83.3 (16.67)
  Role Functioning: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Role Functioning: Final Visit (n=158,161) | 63.5 (2.46) | 68.7 (2.51)
  Emotional Functioning: BL (n=276,287) | 75.4 (1.26) | 73.1 (1.30)
  Emotional Functioning: Week 4 (n=235,250) | 80.5 (1.25) | 77.9 (1.30)
  Emotional Functioning: Week 7 (n=180,220) | 81.3 (1.39) | 80.2 (1.37)
  Emotional Functioning: Week 10 (n=176,202) | 82.9 (1.39) | 81.2 (1.31)
  Emotional Functioning: Week 13 (n=152,183) | 82.6 (1.48) | 80.5 (1.41)
  Emotional Functioning: Week 16 (n=121,165) | 83.1 (1.81) | 81.9 (1.49)
  Emotional Functioning: Week 19 (n=114,143) | 82.2 (1.95) | 82.4 (1.56)
  Emotional Functioning: Week 22 (n=79,143) | 85.9 (2.06) | 84.0 (1.53)
  Emotional Functioning: Week 25 (n=64,124) | 88.2 (1.97) | 84.8 (1.53)
  Emotional Functioning: Week 28 (n=47,111) | 86.0 (2.37) | 85.5 (1.54)
  Emotional Functioning: Week 31 (n=45,95) | 85.7 (2.24) | 85.7 (1.78)
  Emotional Functioning: Week 34 (n=37,87) | 88.5 (2.29) | 85.4 (1.86)
  Emotional Functioning: Week 37 (n=29,64) | 83.9 (3.43) | 86.3 (2.12)
  Emotional Functioning: Week 40 (n=24,55) | 83.6 (3.99) | 86.7 (2.23)
  Emotional Functioning: Week 43 (n=12,43) | 81.9 (5.21) | 87.8 (2.22)
  Emotional Functioning: Week 46 (n=14,42) | 82.1 (4.44) | 87.5 (2.56)
  Emotional Functioning: Week 49 (n=10,36) | 88.3 (4.16) | 91.4 (2.41)
  Emotional Functioning: Week 52 (n=8,29) | 86.5 (5.88) | 88.2 (3.16)
  Emotional Functioning: Week 55 (n=6,24) | 76.4 (9.23) | 88.5 (2.55)
  Emotional Functioning: Week 58 (n=6,21) | 85.6 (6.27) | 88.9 (3.22)
  Emotional Functioning: Week 61 (n=4,17) | 95.8 (2.41) | 90.7 (2.25)
  Emotional Functioning: Week 64 (n=3,20) | 100 (0.00) | 86.3 (3.59)
  Emotional Functioning: Week 67 (n=4,17) | 95.8 (2.41) | 89.2 (3.26)
  Emotional Functioning: Week 70 (n=3,14) | 97.2 (2.78) | 89.3 (4.41)
  Emotional Functioning: Week 73 (n=3,12) | 94.4 (5.56) | 82.9 (5.25)
  Emotional Functioning: Week 76 (n=3,8) | 100.0 (0.00) | 87.5 (6.86)
  Emotional Functioning: Week 79 (n=3,9) | 97.2 (2.78) | 84.3 (7.14)
  Emotional Functioning: Week 82 (n=2,6) | 95.8 (4.17) | 83.3 (13.61)
  Emotional Functioning: Week 85 (n=2,6) | 95.8 (4.17) | 91.7 (5.69)
  Emotional Functioning: Week 88 (n=2,6) | 100.0 (0.00) | 90.3 (3.98)
  Emotional Functioning: Week 91 (n=2,4) | 100.0 (0.00) | 95.8 (4.17)
  Emotional Functioning: Week 94 (n=2,6) | 100.0 (0.00) | 88.9 (5.12)
  Emotional Functioning: Week 97 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 91.7 (5.27)
  Emotional Functioning: Week 100 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 87.5 (4.17)
  Emotional Functioning: Week 103 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 87.5 (5.38)
  Emotional Functioning: Week 106 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 89.6 (3.99)
  Emotional Functioning: Week 109 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 91.7 (4.81)
  Emotional Functioning: Week 112 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.0 (3.33)
  Emotional Functioning: Week 115 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 93.8 (3.99)
  Emotional Functioning: Week 118 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 90.0 (4.86)
  Emotional Functioning: Week 121 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.0 (3.33)
  Emotional Functioning: Week 124 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 90.0 (6.67)
  Emotional Functioning: Week 127 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 100.0 (0.00)
  Emotional Functioning: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 88.9 (11.11)
  Emotional Functioning: Week 133 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 91.7 (8.33)
  Emotional Functioning: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 95.8 (4.17)
  Emotional Functioning: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 95.8 (4.17)
  Emotional Functioning: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 95.8 (4.17)
  Emotional Functioning: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Emotional Functioning: Final Visit (n=158,161) | 75.1 (2.16) | 74.3 (2.00)
  Cognitive Functioning: BL (n=276,287) | 86.9 (1.06) | 85.7 (1.20)
  Cognitive Functioning: Week 4 (n=235,250) | 86.0 (1.14) | 86.3 (1.14)
  Cognitive Functioning: Week 7 (n=180,220) | 85.7 (1.36) | 86.5 (1.24)
  Cognitive Functioning: Week 10 (n=176,202) | 85.6 (1.35) | 86.8 (1.22)
  Cognitive Functioning: Week 13 (n=152,183) | 88.2 (1.34) | 85.7 (1.43)
  Cognitive Functioning: Week 16 (n=121,165) | 82.8 (1.70) | 86.8 (1.48)
  Cognitive Functioning: Week 19 (n=114,143) | 84.2 (1.62) | 87.6 (1.40)
  Cognitive Functioning: Week 22 (n=79,143) | 85.9 (1.92) | 87.4 (1.53)
  Cognitive Functioning: Week 25 (n=64,124) | 85.9 (2.20) | 87.4 (1.50)
  Cognitive Functioning: Week 28 (n=47,111) | 86.5 (2.25) | 88.0 (1.54)
  Cognitive Functioning: Week 31 (n=45,95) | 87.0 (2.18) | 90.0 (1.66)
  Cognitive Functioning: Week 34 (n=37,87) | 88.3 (2.49) | 88.7 (1.69)
  Cognitive Functioning: Week 37 (n=29,64) | 88.5 (2.63) | 91.4 (1.89)
  Cognitive Functioning: Week 40 (n=24,55) | 83.3 (3.48) | 91.5 (1.93)
  Cognitive Functioning: Week 43 (n=12,43) | 88.9 (3.75) | 91.5 (2.10)
  Cognitive Functioning: Week 46 (n=14,42) | 89.3 (3.75) | 91.7 (2.14)
  Cognitive Functioning: Week 49 (n=10,36) | 85.0 (5.80) | 92.6 (2.43)
  Cognitive Functioning: Week 52 (n=8,29) | 91.7 (5.46) | 89.7 (3.35)
  Cognitive Functioning: Week 55 (n=6,24) | 94.4 (5.56) | 91.0 (2.65)
  Cognitive Functioning: Week 58 (n=6,21) | 91.7 (5.69) | 90.5 (3.37)
  Cognitive Functioning: Week 61 (n=4,17) | 91.7 (8.33) | 91.2 (3.53)
  Cognitive Functioning: Week 64 (n=3,20) | 100.0 (0.00) | 93.3 (3.29)
  Cognitive Functioning: Week 67 (n=4,17) | 91.7 (8.33) | 91.2 (4.07)
  Cognitive Functioning: Week 70 (n=3,14) | 100.0 (0.00) | 91.7 (4.19)
  Cognitive Functioning: Week 73 (n=3,12) | 100.0 (0.00) | 83.3 (4.59)
  Cognitive Functioning: Week 76 (n=3,8) | 100.0 (0.00) | 83.3 (8.33)
  Cognitive Functioning: Week 79 (n=3,9) | 100.0 (0.00) | 81.5 (7.58)
  Cognitive Functioning: Week 82 (n=2,6) | 100.0 (0.00) | 88.9 (5.56)
  Cognitive Functioning: Week 85 (n=2,6) | 100.0 (0.00) | 91.7 (5.69)
  Cognitive Functioning: Week 88 (n=2,6) | 100.0 (0.00) | 94.4 (3.51)
  Cognitive Functioning: Week 91 (n=2,4) | 100.0 (0.00) | 95.8 (4.17)
  Cognitive Functioning: Week 94 (n=2,6) | 100.0 (0.00) | 94.4 (3.51)
  Cognitive Functioning: Week 97 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 90.0 (6.67)
  Cognitive Functioning: Week 100 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.8 (4.17)
  Cognitive Functioning: Week 103 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 91.7 (4.81)
  Cognitive Functioning: Week 106 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.8 (4.17)
  Cognitive Functioning: Week 109 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.8 (4.17)
  Cognitive Functioning: Week 112 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 93.3 (4.08)
  Cognitive Functioning: Week 115 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.8 (4.17)
  Cognitive Functioning: Week 118 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.7 (3.33)
  Cognitive Functioning: Week 121 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.7 (3.33)
  Cognitive Functioning: Week 124 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.7 (3.33)
  Cognitive Functioning: Week 127 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 100.0 (0.00)
  Cognitive Functioning: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 88.9 (11.11)
  Cognitive Functioning: Week 133 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 94.4 (5.56)
  Cognitive Functioning: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (0.00)
  Cognitive Functioning: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (0.00)
  Cognitive Functioning: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (0.00)
  Cognitive Functioning: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Cognitive Functioning: Final Visit (n=158,161) | 79.5 (1.82) | 80.0 (2.05)
  Social Functioning: BL (n=276,286) | 72.4 (1.63) | 72.0 (1.77)
  Social Functioning: Week 4 (n=235,250) | 72.1 (1.66) | 74.1 (1.67)
  Social Functioning: Week 7 (n=179,220) | 73.1 (1.88) | 75.1 (1.70)
  Social Functioning: Week 10 (n=176,202) | 74.5 (1.84) | 76.7 (1.65)
  Social Functioning: Week 13 (n=152,183) | 72.7 (2.11) | 76.3 (1.90)
  Social Functioning: Week 16 (n=180,165) | 72.7 (2.52) | 77.5 (1.88)
  Social Functioning: Week 19 (n=114,143) | 74.4 (2.41) | 79.5 (1.93)
  Social Functioning: Week 22 (n=79,143) | 79.3 (2.77) | 80.1 (2.03)
  Social Functioning: Week 25 (n=64,124) | 83.3 (2.43) | 80.2 (1.78)
  Social Functioning: Week 28 (n=47,111) | 83.0 (3.38) | 80.2 (2.05)
  Social Functioning: Week 31 (n=45,95) | 81.5 (3.90) | 78.9 (2.42)
  Social Functioning: Week 34 (n=37,87) | 84.7 (3.06) | 80.7 (2.45)
  Social Functioning: Week 37 (n=29,64) | 85.1 (4.48) | 81.8 (2.59)
  Social Functioning: Week 40 (n=24,55) | 85.4 (4.05) | 82.7 (2.73)
  Social Functioning: Week 43 (n=12,43) | 87.5 (4.64) | 84.1 (2.77)
  Social Functioning: Week 46 (n=14,42) | 86.9 (4.34) | 86.9 (2.70)
  Social Functioning: Week 49 (n=10,36) | 85.0 (5.24) | 84.7 (3.00)
  Social Functioning: Week 52 (n=8,29) | 87.5 (6.10) | 82.2 (3.87)
  Social Functioning: Week 55 (n=6,24) | 86.1 (6.69) | 85.4 (3.80)
  Social Functioning: Week 58 (n=6,21) | 88.9 (5.56) | 87.3 (4.13)
  Social Functioning: Week 61 (n=4,17) | 91.7 (4.81) | 90.2 (3.52)
  Social Functioning: Week 64 (n=3,20) | 94.4 (5.56) | 85.8 (3.68)
  Social Functioning: Week 67 (n=4,17) | 95.8 (4.17) | 85.3 (4.71)
  Social Functioning: Week 70 (n=3,14) | 94.4 (5.56) | 86.9 (4.34)
  Social Functioning: Week 73 (n=3,12) | 100.0 (0.00) | 80.6 (5.36)
  Social Functioning: Week 76 (n=3,8) | 94.4 (5.56) | 81.3 (7.34)
  Social Functioning: Week 79 (n=3,9) | 94.4 (5.56) | 85.2 (7.58)
  Social Functioning: Wek 82 (n=2,6) | 100.0 (0.00) | 80.6 (6.69)
  Social Functioning: Week 85 (n=2,6) | 91.7 (8.33) | 88.9 (7.03)
  Social Functioning: Week 88 (n=2,6) | 91.7 (8.33) | 88.9 (5.56)
  Social Functioning: Week 91 (n=2,4) | 100.0 (0.00) | 91.7 (8.33)
  Social Functioning: Week 94 (n=2,6) | 100.0 (0.00) | 91.7 (5.69)
  Social Functioning: Week 97 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 90.0 (6.67)
  Social Functioning: Week 100 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.8 (4.17)
  Social Functioning: Week 103 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 100.0 (0.00)
  Social Functioning: Week 106 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 91.7 (8.33)
  Social Functioning: Week 109 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.8 (4.17)
  Social Functioning: Week 112 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.7 (3.33)
  Social Functioning: Week 115 (n=1,4) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 95.8 (4.17)
  Social Functioning: Week 118 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.7 (3.33)
  Social Functioning: Week 121 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 100.0 (0.00)
  Social Functioning: Week 124 (n=1,5) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 96.7 (3.33)
  Social Functioning: Week 127 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 83.3 (9.62)
  Social Functioning: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 94.4 (5.56)
  Social Functioning: Week 133 (n=1,3) | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 100.0 (0.00)
  Social Functioning: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (0.00)
  Social Functioning: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (0.00)
  Social Functioning: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (0.00)
  Social Functioning: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 100.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Social Functioning: Final Visit (n=158,161) | 68.1 (2.41) | 71.4 (2.39)
  Fatigue: BL (n=276,287) | 36.3 (1.37) | 34.2 (1.41)
  Fatigue: Week 4 (n=235,250) | 37.1 (1.47) | 34.5 (1.34)
  Fatigue: Week 7 (n=181,220) | 34.4 (1.54) | 34.1 (1.48)
  Fatigue: Week 10 (n=176,201) | 35.3 (1.70) | 33.2 (1.50)
  Fatigue: Week 13 (n=152,183) | 32.9 (1.70) | 33.7 (1.71)
  Fatigue: Week 16 (n=121,165) | 33.0 (2.09) | 32.8 (1.76)
  Fatigue: Week 19 (n=114,143) | 33.1 (2.11) | 29.4 (1.87)
  Fatigue: Week 22 (n=79,143) | 30.0 (2.63) | 26.7 (1.76)
  Fatigue: Week 25 (n=64,124) | 22.2 (2.55) | 25.1 (1.90)
  Fatigue: Week 28 (n=47,110) | 24.1 (3.16) | 23.2 (1.93)
  Fatigue: Week 31 (n=45,95) | 22.0 (2.92) | 22.2 (2.17)
  Fatigue: Week 34 (n=37,87) | 22.8 (3.63) | 19.7 (2.28)
  Fatigue: Week 37 (n=29,64) | 21.8 (4.63) | 19.8 (2.52)
  Fatigue: Week 40 (n=24,55) | 23.6 (4.45) | 18.6 (2.33)
  Fatigue: Week 43 (n=12,43) | 19.4 (3.90) | 17.1 (2.68)
  Fatigue: Week 46 (n=14,42) | 20.6 (4.18) | 13.8 (2.36)
  Fatigue: Week 49 (n=10,36) | 19.4 (3.23) | 14.5 (2.38)
  Fatigue: Week 52 (n=8,30) | 16.7 (2.97) | 17.2 (3.48)
  Fatigue: Week 55 (n=6,24) | 18.5 (5.49) | 14.4 (3.75)
  Fatigue: Week 58 (n=6,21) | 16.7 (4.76) | 16.4 (3.22)
  Fatigue: Week 61 (n=4,17) | 8.3 (5.32) | 14.4 (3.53)
  Fatigue: Week 64 (n=3,20) | 7.4 (3.70) | 17.2 (4.15)
  Fatigue: Week 67 (n=4,17) | 13.9 (2.78) | 15.0 (4.04)
  Fatigue: Week 70 (n=3,14) | 11.1 (0.00) | 16.7 (5.04)
  Fatigue: Week 73 (n=3,12) | 7.4 (3.70) | 16.7 (5.38)
  Fatigue: Week 76 (n=3,8) | 7.4 (3.70) | 18.1 (6.94)
  Fatigue: Week 79 (n=3,9) | 7.4 (3.70) | 18.5 (7.64)
  Fatigue: Week 82 (n=2,6) | 0.0 (0.00) | 29.6 (8.92)
  Fatigue: Week 85 (n=2,6) | 5.6 (5.56) | 11.1 (5.74)
  Fatigue: Week 88 (n=2,6) | 0.0 (0.00) | 9.3 (3.41)
  Fatigue: Week 91 (n=2,4) | 0.0 (0.00) | 11.1 (7.86)
  Fatigue: Week 94 (n=2,6) | 0.0 (0.00) | 7.4 (5.49)
  Fatigue: Week 97 (n=1,5) | 11.1 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (6.09)
  Fatigue: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (7.86)
  Fatigue: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 19.4 (5.32)
  Fatigue: Week 106 (n=1,4) | 11.1 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 13.9 (6.99)
  Fatigue: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (7.17)
  Fatigue: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 17.8 (6.67)
  Fatigue: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 25.0 (5.32)
  Fatigue: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 17.8 (6.67)
  Fatigue: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 17.8 (6.67)
  Fatigue: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 13.3 (6.48)
  Fatigue: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 14.8 (9.80)
  Fatigue: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 18.5 (7.41)
  Fatigue: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 14.8 (9.80)
  Fatigue: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 22.2 (11.11)
  Fatigue: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 22.2 (11.11)
  Fatigue: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 22.2 (11.11)
  Fatigue: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 11.1 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Fatigue: Final Visit (n=158,160) | 40.4 (2.17) | 37.6 (2.31)
  Nausea & Vomiting: BL (n=276,287) | 15.0 (1.39) | 15.7 (1.36)
  Nausea & Vomiting: Week 4 (n=235,250) | 16.6 (1.45) | 19.7 (1.46)
  Nausea & Vomiting: Week 7 (n=181,220) | 16.9 (1.66) | 18.9 (1.63)
  Nausea & Vomiting: Week 10 (n=176,201) | 16.4 (1.67) | 16.4 (1.56)
  Nausea & Vomiting: Week 13 (n=121,183) | 12.8 (1.41) | 14.7 (1.55)
  Nausea & Vomiting: Week 16 (n=121,165) | 14.2 (1.99) | 14.5 (1.56)
  Nausea & Vomiting: Week 19 (n=114,143) | 14.2 (2.01) | 13.9 (1.59)
  Nausea & Vomiting: Week 22 (n=79,143) | 10.3 (2.23) | 12.2 (1.66)
  Nausea & Vomiting: Week 25 (n=64,124) | 8.6 (2.38) | 8.2 (1.48)
  Nausea & Vomiting: Week 28 (n=47,110) | 3.5 (1.34) | 6.5 (1.52)
  Nausea & Vomiting: Week 31 (n=45,95) | 3.7 (1.58) | 8.8 (2.02)
  Nausea & Vomiting: Week 34 (n=37,87) | 4.5 (1.90) | 7.5 (1.90)
  Nausea & Vomiting: Week 37 (n=29,64) | 2.9 (1.67) | 6.8 (2.34)
  Nausea & Vomiting: Week 40 (n=24,55) | 4.2 (1.50) | 4.8 (1.87)
  Nausea & Vomiting: Week 43 (n=12,43) | 2.8 (1.87) | 1.2 (0.66)
  Nausea & Vomiting: Week 46 (n=14,42) | 1.2 (1.19) | 2.8 (1.12)
  Nausea & Vomiting: Week 49 (n=10,36) | 3.3 (2.22) | 0.9 (0.65)
  Nausea & Vomiting: Week 52 (n=8,30) | 2.1 (2.08) | 5.0 (2.90)
  Nausea & Vomiting: Week 55 (n=6,24) | 0.0 (0.00) | 2.1 (1.15)
  Nausea & Vomiting: Week 58 (n=6,21) | 0.0 (0.00) | 3.2 (2.19)
  Nausea & Vomiting: Week 61 (n=4,17) | 0.0 (0.00) | 0.0 (0.00)
  Nausea & Vomiting: Week 64 (n=3,20) | 0.0 (0.00) | 4.2 (2.38)
  Nausea & Vomiting: Week 67 (n=4,17) | 0.0 (0.00) | 2.9 (2.14)
  Nausea & Vomiting: Week 70 (n=3,14) | 0.0 (0.00) | 2.4 (2.38)
  Nausea & Vomiting: Week 73 (n=3,12) | 0.0 (0.00) | 1.4 (1.39)
  Nausea & Vomiting: Week 76 (n=3,8) | 5.6 (5.56) | 0.0 (0.00)
  Nausea & Vomiting: Week 79 (n=3,9) | 0.0 (0.00) | 0.0 (0.00)
  Nausea & Vomiting: Week 82 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Nausea & Vomiting: Week 85 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Nausea & Vomiting: Week 88 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Nausea & Vomiting: Week 91 (n=2,4) | 0.0 (0.00) | 0.0 (0.00)
  Nausea & Vomiting: Week 94 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Nausea & Vomiting: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Nausea & Vomiting: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Nausea & Vomiting: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Nausea & Vomiting: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Nausea & Vomiting: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Nausea & Vomiting: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Nausea & Vomiting: Final Visit (n=158,161) | 14.9 (1.79) | 19.8 (2.36)
  Pain: BL (n=276,287) | 24.9 (1.46) | 25.1 (1.55)
  Pain: Week 4 (n=235,250) | 17.8 (1.43) | 17.9 (1.30)
  Pain: Week 7 (n=181,220) | 14.5 (1.43) | 16.1 (1.50)
  Pain: Week 10 (n=176,202) | 13.4 (1.34) | 14.4 (1.42)
  Pain: Week 13 (n=152,183) | 12.0 (1.42) | 13.3 (1.45)
  Pain: Week 16 (n=121,165) | 13.6 (1.80) | 12.4 (1.54)
  Pain: Week 19 (n=114,143) | 14.2 (1.98) | 12.8 (1.68)
  Pain: Week 22 (n=79,143) | 15.0 (2.59) | 13.2 (1.80)
  Pain: Week 25 (n=64,124) | 10.7 (2.44) | 12.2 (1.90)
  Pain: Week 28 (n=47,111) | 8.2 (1.82) | 12.0 (1.97)
  Pain: Week 31 (n=45,95) | 12.2 (2.97) | 11.8 (2.22)
  Pain: Week 34 (n=37,87) | 12.2 (3.00) | 11.3 (2.32)
  Pain: Week 37 (n=29,64) | 11.5 (2.99) | 12.2 (2.90)
  Pain: Week 40 (n=24,55) | 18.8 (4.74) | 10.3 (2.75)
  Pain: Week 43 (n=12,43) | 16.7 (5.03) | 8.9 (2.44)
  Pain: Week 46 (n=14,42) | 13.1 (3.57) | 6.7 (2.48)
  Pain: Week 49 (n=10,36) | 13.3 (4.84) | 6.5 (2.23)
  Pain: Week 52 (n=8,30) | 6.3 (3.05) | 10.0 (4.49)
  Pain: Week 55 (n=6,24) | 2.8 (2.78) | 8.3 (4.01)
  Pain: Week 58 (n=6,21) | 8.3 (5.69) | 7.1 (3.56)
  Pain: Week 61 (n=4,17) | 0.0 (0.00) | 4.9 (3.43)
  Pain: Week 64 (n=3,20) | 5.6 (5.56) | 6.7 (3.06)
  Pain: Week 67 (n=4,17) | 0.0 (0.00) | 4.9 (2.77)
  Pain: Week 70 (n=3,14) | 0.0 (0.00) | 4.8 (4.76)
  Pain: Week 73 (n=3,12) | 5.6 (5.56) | 9.7 (5.97)
  Pain: Week 76 (n=3,8) | 5.6 (5.56) | 8.3 (8.33)
  Pain: Week 79 (n=3,9) | 5.6 (5.56) | 9.3 (7.41)
  Pain: Week 82 (n=2,6) | 0.0 (0.00) | 2.8 (2.78)
  Pain: Week 85 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Pain: Week 88 (n=2,6) | 0.0 (0.00) | 2.8 (2.78)
  Pain: Week 91 (n=2,4) | 0.0 (0.00) | 4.2 (4.17)
  Pain: Week 94 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Pain: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 3.3 (3.33)
  Pain: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Pain: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Pain: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Pain: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Pain: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 3.3 (3.33)
  Pain: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Pain: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 3.3 (3.33)
  Pain: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 3.3 (3.33)
  Pain: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Pain: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Pain: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 5.6 (5.56)
  Pain: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 5.6 (5.56)
  Pain: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Pain: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Pain: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Pain: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Pain: Final Visit (n=158,161) | 27.4 (2.34) | 25.4 (2.49)
  Dyspnoea: BL (n=274,281) | 12.4 (1.25) | 13.4 (1.23)
  Dyspnoea: Week 4 (n=232,249) | 12.1 (1.35) | 11.8 (1.24)
  Dyspnoea: Week 7 (n=181,217) | 12.7 (1.66) | 10.8 (1.21)
  Dyspnoea: Week 10 (n=176,198) | 14.6 (1.71) | 11.3 (1.33)
  Dyspnoea: Week 13 (n=151,182) | 11.3 (1.80) | 13.7 (1.74)
  Dyspnoea: Week 16 (n=121,165) | 15.4 (2.28) | 13.5 (1.79)
  Dyspnoea: Week 19 (n=113,143) | 15.3 (2.48) | 11.9 (1.70)
  Dyspnoea: Week 22 (n=79,143) | 13.9 (2.79) | 12.1 (1.64)
  Dyspnoea: Week 25 (n=63,124) | 12.7 (2.76) | 9.4 (1.60)
  Dyspnoea: Week 28 (n=47,110) | 9.2 (2.42) | 10.3 (1.76)
  Dyspnoea: Week 31 (n=45,95) | 10.4 (2.56) | 9.1 (1.69)
  Dyspnoea: Week 34 (n=36,87) | 10.2 (2.92) | 9.6 (2.10)
  Dyspnoea: Week 37 (n=29,64) | 10.3 (3.35) | 10.4 (2.45)
  Dyspnoea: Week 40 (n=24,55) | 9.7 (3.74) | 4.8 (1.60)
  Dyspnoea: Week 43 (n=12,43) | 19.4 (7.63) | 6.2 (2.00)
  Dyspnoea: Week 46 (n=14,42) | 11.9 (4.43) | 5.6 (1.94)
  Dyspnoea: Week 49 (n=10,36) | 6.7 (4.44) | 4.6 (1.95)
  Dyspnoea: Week 52 (n=8,30) | 12.5 (6.10) | 5.6 (2.31)
  Dyspnoea: Week 55 (n=6,24) | 5.6 (5.56) | 8.3 (3.01)
  Dyspnoea: Week 58 (n=6,21) | 5.6 (5.56) | 6.3 (3.72)
  Dyspnoea: Week 61 (n=4,17) | 16.7 (9.62) | 3.9 (2.68)
  Dyspnoea: Week 64 (n=3,20) | 0.0 (0.00) | 8.3 (4.10)
  Dyspnoea: Week 67 (n=4,17) | 8.3 (8.33) | 5.9 (4.27)
  Dyspnoea: Week 70 (n=3,14) | 0.0 (0.00) | 7.1 (5.16)
  Dyspnoea: Week 73 (n=3,12) | 0.0 (0.00) | 8.3 (4.35)
  Dyspnoea: Week 76 (n=3,8) | 11.1 (11.11) | 8.3 (5.46)
  Dyspnoea: Week 79 (n=3,9) | 0.0 (0.00) | 7.4 (4.90)
  Dyspnoea: Week 82 (n=2,6) | 0.0 (0.00) | 16.7 (11.39)
  Dyspnoea: Week 85 (n=180,6) | 0.0 (0.00) | 5.6 (5.56)
  Dyspnoea: Week 88 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Dyspnoea: Week 91 (n=2,4) | 0.0 (0.00) | 8.3 (8.33)
  Dyspnoea: Week 94 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Dyspnoea: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dyspnoea: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dyspnoea: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Dyspnoea: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Dyspnoea: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Dyspnoea: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Dyspnoea: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Dyspnoea: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Dyspnoea: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Dyspnoea: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Dyspnoea: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (11.11)
  Dyspnoea: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 11.1 (11.11)
  Dyspnoea: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (11.11)
  Dyspnoea: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 16.7 (16.67)
  Dyspnoea: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 16.7 (16.67)
  Dyspnoea: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 16.7 (16.67)
  Dyspnoea: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 33.3 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Dyspnoea: Final Visit (n=157,160) | 20.0 (2.13) | 18.3 (2.11)
  Insomnia: BL (n=276,285) | 27.2 (1.86) | 23.6 (1.71)
  Insomnia: Week 4 (n=234,248) | 22.1 (1.82) | 23.3 (1.65)
  Insomnia: Week 7 (n=181,219) | 21.9 (2.10) | 20.4 (1.69)
  Insomnia: Week 10 (n=175,200) | 19.8 (2.04) | 18.0 (1.63)
  Insomnia: Week 13 (n=152,183) | 14.7 (1.86) | 18.9 (1.70)
  Insomnia: Week 16 (n=120,164) | 15.3 (1.93) | 17.7 (1.88)
  Insomnia: Week 19 (n=113,143) | 17.1 (2.30) | 20.0 (2.10)
  Insomnia: Week 22 (n=79,143) | 14.8 (2.38) | 17.0 (2.24)
  Insomnia: Week 25 (n=64,124) | 15.1 (3.05) | 15.9 (2.14)
  Insomnia: Week 28 (n=47,110) | 9.9 (3.03) | 13.3 (2.07)
  Insomnia: Week 31 (n=45,94) | 10.4 (2.77) | 14.9 (2.34)
  Insomnia: Week 34 (n=37,87) | 9.0 (2.78) | 13.4 (2.07)
  Insomnia: Week 37 (n=29,63) | 8.0 (3.16) | 11.1 (2.26)
  Insomnia: Week 40 (n=24,55) | 13.9 (4.45) | 10.3 (2.58)
  Insomnia: Week 43 (n=12,43) | 13.9 (8.66) | 9.3 (2.79)
  Insomnia: Week 46 (n=13,42) | 7.7 (4.05) | 9.5 (2.85)
  Insomnia: Week 49 (n=10,36) | 10.0 (7.11) | 7.4 (2.69)
  Insomnia: Week 52 (n=8,30) | 12.5 (6.10) | 7.8 (3.07)
  Insomnia: Week 55 (n=6,24) | 16.7 (7.45) | 8.3 (3.01)
  Insomnia: Week 58 (n=6,21) | 11.1 (7.03) | 9.5 (4.08)
  Insomnia: Week 61 (n=4,17) | 8.3 (8.33) | 7.8 (4.55)
  Insomnia: Week 64 (n=3,20) | 0.0 (0.00) | 10.0 (4.90)
  Insomnia: Week 67 (n=4,17) | 0.0 (0.00) | 9.8 (4.75)
  Insomnia: Week 70 (n=3,14) | 0.0 (0.00) | 9.5 (5.45)
  Insomnia: Week 73 (n=3,12) | 0.0 (0.00) | 11.1 (6.27)
  Insomnia: Week 76 (n=3,8) | 0.0 (0.00) | 8.3 (5.46)
  Insomnia: Week 79 (n=3,9) | 0.0 (0.00) | 11.1 (5.56)
  Insomnia: Week 82 (n=2,6) | 0.0 (0.00) | 11.1 (11.11)
  Insomnia: Week 85 (n=2,6) | 0.0 (0.00) | 11.1 (7.03)
  Insomnia: Week 88 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Insomnia: Week 91 (n=2,4) | 0.0 (0.00) | 0.0 (0.00)
  Insomnia: Week 94 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Insomnia: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Insomnia: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Insomnia: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Insomnia: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Insomnia: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Insomnia: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Insomnia: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Insomnia: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Insomnia: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Insomnia: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Insomnia: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Insomnia: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 11.1 (11.11)
  Insomnia: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (11.11)
  Insomnia: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Insomnia: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Insomnia: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Insomnia: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Insomnia: Final Visit (n=157,160) | 21.9 (2.29) | 24.6 (2.28)
  Appetite Loss: BL (n=275,286) | 35.2 (2.02) | 33.8 (2.04)
  Appetite Loss: Week 4 (n=235,250) | 31.5 (2.01) | 33.6 (2.01)
  Appetite Loss: Week 7 (n=180,216) | 27.2 (2.19) | 31.3 (2.04)
  Appetite Loss: Week 10 (n=176,201) | 26.7 (2.10) | 29.4 (2.08)
  Appetite Loss: Week 13 (n=151,183) | 24.7 (2.11) | 28.4 (2.17)
  Appetite Loss: Week 16 (n=121,165) | 24.5 (2.27) | 27.9 (2.23)
  Appetite Loss: Week 19 (n=114,141) | 26.9 (2.81) | 25.1 (2.40)
  Appetite Loss: Week 22 (n=79,143) | 19.0 (2.92) | 20.7 (2.19)
  Appetite Loss: Week 25 (n=64,124) | 12.0 (2.39) | 16.7 (1.96)
  Appetite Loss: Week 28 (n=47,109) | 14.2 (2.82) | 11.6 (1.96)
  Appetite Loss: Week 31 (n=45,95) | 11.1 (3.18) | 13.0 (2.61)
  Appetite Loss: Week 34 (n=37,87) | 11.7 (2.65) | 9.6 (2.24)
  Appetite Loss: Week 37 (n=29,64) | 12.6 (3.48) | 10.9 (2.78)
  Appetite Loss: Week 40 (n=24,55) | 13.9 (3.97) | 9.7 (2.69)
  Appetite Loss: Week 43 (n=12,43) | 5.6 (3.75) | 7.0 (2.37)
  Appetite Loss: Week 46 (n=14,42) | 4.8 (3.24) | 5.6 (2.25)
  Appetite Loss: Week 49 (n=9,36) | 3.7 (3.70) | 6.5 (2.23)
  Appetite Loss: Week 52 (n=8,30) | 0.0 (0.00) | 10.0 (3.96)
  Appetite Loss: Week 55 (n=6,24) | 0.0 (0.00) | 10.0 (3.96)
  Appetite Loss: Week 58 (n=6,21) | 5.6 (5.56) | 4.8 (2.61)
  Appetite Loss: Week 61 (n=4,17) | 8.3 (8.33) | 0.0 (0.00)
  Appetite Loss: Week 64 (n=3,20) | 0.0 (0.00) | 8.3 (4.10)
  Appetite Loss: Week 67 (n=4,17) | 8.3 (8.33) | 5.9 (3.18)
  Appetite Loss: Week 70 (n=3,14) | 0.0 (0.00) | 7.1 (5.16)
  Appetite Loss: Week 73 (n=3,12) | 0.0 (0.00) | 5.6 (3.75)
  Appetite Loss: Week 76 (n=3,8) | 0.0 (0.00) | 4.2 (4.17)
  Appetite Loss: Week 79 (n=3,9) | 0.0 (0.00) | 0.0 (0.00)
  Appetite Loss: Week 82 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Appetite Loss: Week 85 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Appetite Loss: Week 88 (n=2,6) | 0.0 (0.00) | 11.1 (7.03)
  Appetite Loss: Week 91 (n=2,4) | 0.0 (0.00) | 0.0 (0.00)
  Appetite Loss: Week 94 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Appetite Loss: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Appetite Loss: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Appetite Loss: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Appetite Loss: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 11.1 (11.11)
  Appetite Loss: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (11.11)
  Appetite Loss: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Appetite Loss: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Appetite Loss: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Appetite Loss: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Appetite Loss: Week Final Visit (n=156,161) | 35.3 (2.45) | 33.5 (2.76)
  Constipation: BL (n=276,285) | 22.9 (1.79) | 21.5 (1.69)
  Constipation: Week 4 (n=235,247) | 20.6 (1.85) | 20.2 (1.76)
  Constipation: Week 7 (n=179,220) | 19.0 (2.01) | 17.6 (1.79)
  Constipation: Week 10 (n=175,203) | 19.2 (1.90) | 15.1 (1.68)
  Constipation: Week 13 (n=152,183) | 16.7 (1.92) | 15.8 (1.73)
  Constipation: Week 16 (n=121,165) | 14.6 (1.99) | 15.4 (1.87)
  Constipation: Week 19 (n=114,143) | 13.5 (2.11) | 14.5 (1.94)
  Constipation: Week 22 (n=78,143) | 12.0 (2.27) | 10.0 (1.62)
  Constipation: Week 25 (n=64,124) | 7.3 (2.40) | 10.2 (1.71)
  Constipation: Week 28 (n=47,111) | 7.8 (2.31) | 9.6 (1.93)
  Constipation: Week 31 (n=45,95) | 10.4 (2.96) | 6.3 (1.68)
  Constipation: Week 34 (n=37,86) | 5.4 (2.05) | 4.7 (1.48)
  Constipation: Week 37 (n=29,64) | 11.5 (3.80) | 10.4 (2.96)
  Constipation: Week 40 (n=24,55) | 8.3 (3.62) | 7.9 (2.28)
  Constipation: Week 43 (n=12,43) | 8.3 (4.35) | 7.0 (2.37)
  Constipation: Week 46 (n=14,42) | 4.8 (3.24) | 7.1 (2.90)
  Constipation: Week 49 (n=10,36) | 3.3 (3.33) | 5.6 (2.10)
  Constipation: Week 52 (n=8,29) | 4.2 (4.17) | 10.3 (4.09)
  Constipation: Week 55 (n=6,24) | 5.6 (5.56) | 6.9 (4.48)
  Constipation: Week 58 (n=6,21) | 11.1 (7.03) | 6.3 (3.72)
  Constipation: Week 61 (n=4,17) | 8.3 (8.33) | 5.9 (4.27)
  Constipation: Week 64 (n=3,20) | 0.0 (0.00) | 5.0 (3.65)
  Constipation: Week 67 (n=4,17) | 0.0 (0.00) | 5.9 (4.27)
  Constipation: Week 70 (n=3,14) | 0.0 (0.00) | 4.8 (4.76)
  Constipation: Week 73 (n=3,12) | 0.0 (0.00) | 11.1 (6.27)
  Constipation: Week 76 (n=3,8) | 0.0 (0.00) | 4.2 (4.17)
  Constipation: Week 79 (n=3,9) | 0.0 (0.00) | 3.7 (3.70)
  Constipation: Week 82 (n=2,6) | 16.7 (16.67) | 16.7 (16.67)
  Constipation: Week 85 (n=2,6) | 16.7 (16.67) | 0.0 (0.00)
  Constipation: Week 88 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Constipation: Week 91 (n=2,4) | 0.0 (0.00) | 0.0 (0.00)
  Constipation: Week 94 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Constipation: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Constipation: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Constipation: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Constipation: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Constipation: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Constipation: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Constipation: Final Visit (n=158,160) | 19.0 (2.12) | 20.0 (2.16)
  Diarrhoea: BL (n=276,283) | 10.9 (1.21) | 10.7 (1.14)
  Diarrhoea: Week 4 (n=234,246) | 9.1 (1.25) | 12.2 (1.30)
  Diarrhoea: Week 7 (n=180,220) | 8.7 (1.40) | 14.2 (1.65)
  Diarrhoea: Week 10 (n=174,202) | 10.5 (1.51) | 11.9 (1.55)
  Diarrhoea: Week 13 (n=152,183) | 6.6 (1.21) | 12.0 (1.66)
  Diarrhoea: Week 16 (n=120,165) | 8.1 (1.63) | 12.9 (1.61)
  Diarrhoea: Week 19 (n=114,143) | 7.3 (1.70) | 10.3 (1.45)
  Diarrhoea: Week 22 (n=78,143) | 6.0 (1.80) | 9.6 (1.43)
  Diarrhoea: Week 25 (n=64,124) | 7.3 (1.74) | 6.2 (1.23)
  Diarrhoea: Week 28 (n=47,111) | 5.7 (1.85) | 4.8 (1.20)
  Diarrhoea: Week 31 (n=45,95) | 5.9 (1.92) | 4.9 (1.32)
  Diarrhoea: Week 34 (n=37,87) | 5.4 (2.05) | 5.7 (1.56)
  Diarrhoea: Week 37 (n=29,64) | 5.7 (2.38) | 4.2 (1.39)
  Diarrhoea: Week 40 (n=24,55) | 6.9 (2.82) | 3.0 (1.79)
  Diarrhoea: Week 43 (n=12,42) | 8.3 (4.35) | 2.4 (1.76)
  Diarrhoea: Week 46 (n=14,42) | 4.8 (3.24) | 1.6 (1.11)
  Diarrhoea: Week 49 (n=10,36) | 10.0 (5.09) | 3.7 (1.77)
  Diarrhoea: Week 52 (n=8,29) | 8.3 (5.46) | 2.3 (1.60)
  Diarrhoea: Week 55 (n=6,24) | 11.1 (7.03) | 4.2 (2.30)
  Diarrhoea: Week 58 (n=6,21) | 11.1 (7.03) | 4.8 (2.61)
  Diarrhoea: Week 61 (n=4,17) | 16.7 (9.62) | 0.0 (0.00)
  Diarrhoea: Week 64 (n=3,20) | 11.1 (11.11) | 3.3 (2.29)
  Diarrhoea: Week 67 (n=4,17) | 16.7 (9.62) | 2.0 (1.96)
  Diarrhoea: Week 70 (n=3,14) | 11.1 (11.11) | 3.3 (2.29)
  Diarrhoea: Week 73 (n=3,12) | 11.1 (11.11) | 2.0 (1.96)
  Diarrhoea: Week 76 (n=3,8) | 22.2 (11.11) | 0.0 (0.00)
  Diarrhoea: Week 79 (n=3,9) | 11.1 (11.11) | 0.0 (0.00)
  Diarrhoea: Week 82 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Diarrhoea: Week 85 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Diarrhoea: Week 88 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Diarrhoea: Week 91 (n=2,4) | 16.7 (16.67) | 0.0 (0.00)
  Diarrhoea: Week 94 (n=2,6) | 16.7 (16.67) | 0.0 (0.00)
  Diarrhoea: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Diarrhoea: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Diarrhoea: Week 127 (n=1,3) | 0.0 (0) | 0.0 (0.00)
  Diarrhoea: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Diarrhoea: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Diarrhoea: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Diarrhoea: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Diarrhoea: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Diarrhoea: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Diarrhoea: Final Visit (n=157,160) | 10.0 (1.55) | 10.0 (1.67)
  Financial Difficulties: BL (n=274,286) | 27.3 (1.91) | 29.3 (1.89)
  Financial Difficulties: Week 4 (n=234,249) | 23.6 (1.93) | 27.7 (1.99)
  Financial Difficulties: Week 7 (n=178,220) | 23.6 (2.08) | 23.9 (1.96)
  Financial Difficulties: Week 10 (n=175,202) | 21.5 (2.11) | 23.3 (2.03)
  Financial Difficulties: Week 13 (n=151,181) | 22.5 (2.23) | 22.7 (2.08)
  Financial Difficulties: Week 16 (n=120,165) | 23.1 (2.58) | 24.4 (2.26)
  Financial Difficulties: Week 19 (n=113,143) | 20.6 (2.53) | 22.4 (2.49)
  Financial Difficulties: Week 22 (n=78,142) | 19.7 (3.01) | 24.9 (2.52)
  Financial Difficulties: Week 25 (n=63,124) | 16.4 (3.01) | 22.3 (2.34)
  Financial Difficulties: Week 28 (n=45,111) | 17.0 (3.76) | 21.6 (2.55)
  Financial Difficulties: Week 31 (n=45,94) | 15.6 (3.76) | 23.4 (2.89)
  Financial Difficulties: Week 34 (n=36,87) | 10.2 (2.92) | 24.5 (2.96)
  Financial Difficulties: Week 37 (n=29,64) | 13.8 (4.83) | 23.4 (3.38)
  Financial Difficulties: Week 40 (n=24,55) | 22.2 (5.18) | 23.6 (3.74)
  Financial Difficulties: Week 43 (n=12,43) | 16.7 (7.68) | 19.4 (3.72)
  Financial Difficulties: Week 46 (n=14,42) | 16.7 (5.79) | 18.3 (3.45)
  Financial Difficulties: Week 49 (n=10,35) | 16.7 (5.56) | 20.0 (4.14)
  Financial Difficulties: Week 52 (n=8,29) | 8.3 (5.46) | 20.7 (4.50)
  Financial Difficulties: Week 55 (n=6,24) | 16.7 (11.39) | 18.1 (5.30)
  Financial Difficulties: Week 58 (n=6,21) | 11.1 (7.03) | 22.2 (6.23)
  Financial Difficulties: Week 61 (n=4,17) | 16.7 (9.62) | 23.5 (6.86)
  Financial Difficulties: Week 64 (n=3,20) | 11.1 (11.11) | 16.7 (4.52)
  Financial Difficulties: Week 67 (n=4,17) | 16.7 (9.62) | 17.6 (5.05)
  Financial Difficulties: Week 70 (n=3,14) | 11.1 (11.11) | 19.0 (5.76)
  Financial Difficulties: Week 73 (n=3,12) | 11.1 (11.11) | 19.4 (4.95)
  Financial Difficulties: Week 76 (n=3,8) | 11.1 (11.11) | 25.0 (8.33)
  Financial Difficulties: Week 79 (n=3,9) | 11.1 (11.11) | 25.9 (10.80)
  Financial Difficulties: Week 82 (n=2,6) | 16.7 (16.67) | 22.2 (7.03)
  Financial Difficulties: Week 85 (n=2,6) | 16.7 (16.67) | 16.7 (7.45)
  Financial Difficulties: Week 88 (n=2,6) | 16.7 (16.67) | 16.7 (7.45)
  Financial Difficulties: Week 91 (n=2,4) | 16.7 (16.67) | 25.0 (8.33)
  Financial Difficulties: Week 94 (n=2,6) | 16.7 (16.67) | 16.7 (7.45)
  Financial Difficulties: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 20.0 (8.16)
  Financial Difficulties: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (9.62)
  Financial Difficulties: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Financial Difficulties: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (9.62)
  Financial Difficulties: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (9.62)
  Financial Difficulties: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 13.3 (8.16)
  Financial Difficulties: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (9.62)
  Financial Difficulties: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 13.3 (8.16)
  Financial Difficulties: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 13.3 (8.16)
  Financial Difficulties: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 13.3 (8.16)
  Financial Difficulties: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (11.11)
  Financial Difficulties: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 11.1 (11.11)
  Financial Difficulties: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Financial Difficulties: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Financial Difficulties: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Financial Difficulties: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (0.00)
  Financial Difficulties: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group at this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Financial Difficulties: Final Visit (n=158,160) | 26.6 (2.39) | 27.9 (2.51)

12. Secondary Outcome: EORTC Quality of Life Questionnaire-Stomach Cancer Specific (QLQ STO22) Questionnaire Scores
Description: The QLQ-STO22 is a gastric cancer quality of life questionnaire. There are 22 questions concerning disease, treatment related symptoms, side effects, dysphagia, nutritional aspects, and questions about the emotional problems of gastric cancer (dysphagia, pain, reflux, eating restrictions, anxiety, dry mouth, body image, and hair loss). The questions are grouped into five scales and 4 single items which are related to the symptoms of the disease. Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100; higher score=better level of functioning or greater degree of symptoms.
Time Frame: as for outcome 11
Population: FAS; n = number of participants assessed for a specific parameter at a given visit.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
scores on a scale
  Dysphagia Scale: BL (n=276,287) | 18.7 (1.27) | 16.6 (1.21)
  Dysphagia Scale: Week 4 (n=234,250) | 11.8 (0.92) | 12.5 (1.01)
  Dysphagia Scale: Week 7 (n=181,220) | 10.9 (1.16) | 12.8 (1.22)
  Dysphagia Scale: Week 10 (n=176,203) | 8.5 (0.97) | 10.6 (1.19)
  Dysphagia Scale: Week 13 (n=152,183) | 8.8 (1.15) | 9.0 (1.09)
  Dysphagia Scale: Week 16 (n=120,165) | 10.2 (1.50) | 9.1 (1.09)
  Dysphagia Scale: Week 19 (n=114,143) | 9.5 (1.52) | 8.8 (1.26)
  Dysphagia Scale: Week 22 (n=79,143) | 10.0 (2.11) | 7.8 (1.19)
  Dysphagia Scale: Week 25 (n=64,124) | 6.9 (1.99) | 6.8 (1.27)
  Dysphagia Scale: Week 28 (n=47,111) | 6.6 (1.84) | 5.3 (1.03)
  Dysphagia Scale: Week 31 (n=45,95) | 6.4 (2.16) | 6.8 (1.40)
  Dysphagia Scale: Week 34 (n=37,87) | 3.9 (1.44) | 7.5 (1.51)
  Dysphagia Scale: Week 37 (n=29,64) | 5.4 (2.04) | 7.3 (2.03)
  Dysphagia Scale: Week 40 (n=24,55) | 3.7 (1.59) | 6.5 (1.82)
  Dysphagia Scale: Week 43 (n=12,43) | 4.6 (2.89) | 5.2 (1.63)
  Dysphagia Scale: Week 46 (n=14,42) | 2.4 (1.26) | 2.9 (1.08)
  Dysphagia Scale: Week 49 (n=10,36) | 4.4 (2.46) | 2.2 (0.74)
  Dysphagia Scale: Week 52 (n=8,30) | 1.4 (1.39) | 4.4 (1.81)
  Dysphagia Scale: Week 55 (n=6,24) | 0.0 (0.00) | 3.7 (1.28)
  Dysphagia Scale: Week 58 (n=6,21) | 3.7 (2.34) | 3.2 (1.56)
  Dysphagia Scale: Week 61 (n=4,17) | 2.8 (2.78) | 0.7 (0.65)
  Dysphagia Scale: Week 64 (n=3,20) | 0.0 (0.00) | 3.3 (1.99)
  Dysphagia Scale: Week 67 (n=4,16) | 2.8 (2.78) | 2.8 (2.15)
  Dysphagia Scale: Week 70 (n=3,14) | 0.0 (0.00) | 3.2 (2.45)
  Dysphagia Scale: Week 73 (n=3,12) | 0.0 (0.00) | 4.6 (2.54)
  Dysphagia Scale: Week 76 (n=3,8) | 0.0 (0.00) | 2.8 (1.82)
  Dysphagia Scale: Week 79 (n=3,9) | 0.0 (0.00) | 2.5 (1.63)
  Dysphagia Scale: Week 82 (n=2,6) | 0.0 (0.00) | 3.7 (2.34)
  Dysphagia Scale: Week 85 (n=2,6) | 0.0 (0.00) | 1.9 (1.85)
  Dysphagia Scale: Week 88 (n=2,6) | 0.0 (0.00) | 1.9 (1.85)
  Dysphagia Scale: Week 91 (n=2,4) | 0.0 (0.00) | 0.0 (0.00)
  Dysphagia Scale: Week 94 (n=2,6) | 0.0 (0.00) | 1.9 (1.85)
  Dysphagia Scale: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 2.2 (2.22)
  Dysphagia Scale: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 2.8 (2.78)
  Dysphagia Scale: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 2.2 (2.22)
  Dysphagia Scale: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Dysphagia Scale: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dysphagia Scale: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Dysphagia Scale: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 5.6 (5.56)
  Dysphagia Scale: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 5.6 (5.56)
  Dysphagia Scale: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Dysphagia Scale: Final Visit (n=157,159 | 15.4 (1.77) | 17.0 (1.92)
  Pain Scale: BL (n=276,287) | 29.7 (1.32) | 27.0 (1.20)
  Pain Scale: Week 4 (n=234,250) | 21.6 (1.15) | 21.8 (1.05)
  Pain Scale: Week 7 (n=181,219) | 19.4 (1.26) | 20.1 (1.30)
  Pain Scale: Week 10 (n=176,203) | 17.0 (1.11) | 17.5 (1.14)
  Pain Scale: Week 13 (n=152,183) | 16.0 (1.25) | 16.2 (1.21)
  Pain Scale: Week 16 (n=120,165) | 17.0 (1.45) | 15.9 (1.23)
  Pain Scale: Week 19 (n=114,143) | 19.2 (1.95) | 16.3 (1.32)
  Pain Scale: Week 22 (n=79,143) | 15.8 (2.05) | 15.1 (1.58)
  Pain Scale: Week 25 (n=64,124) | 11.3 (1.82) | 14.4 (1.63)
  Pain Scale: Week 28 (n=47,111) | 11.2 (1.95) | 14.0 (1.64)
  Pain Scale: Week 31 (n=45,95) | 12.6 (2.33) | 14.6 (2.09)
  Pain Scale: Week 34 (n=37,87) | 12.2 (2.18) | 12.5 (2.04)
  Pain Scale: Week 37 (n=29,64) | 13.8 (2.90) | 13.8 (2.63)
  Pain Scale: Week 40 (n=24,55) | 14.9 (2.97) | 11.8 (2.28)
  Pain Scale: Week 43 (n=12,43) | 13.0 (3.41) | 9.7 (1.98)
  Pain Scale: Week 46 (n=14,42) | 15.5 (3.13) | 10.1 (2.35)
  Pain Scale: Week 49 (n=10,36) | 11.7 (4.51) | 9.5 (1.79)
  Pain Scale: Week 52 (n=8,30) | 9.4 (4.00) | 8.6 (2.69)
  Pain Scale: Week 55 (n=6,24) | 9.7 (5.01) | 4.5 (1.42)
  Pain Scale: Week 58 (n=6,21) | 5.6 (4.12) | 6.3 (1.90)
  Pain Scale: Week 61 (n=4,17) | 4.2 (2.41) | 5.4 (2.36)
  Pain Scale: Week 64 (n=3,20) | 2.8 (2.78) | 9.6 (2.28)
  Pain Scale: Week 67 (n=4,16) | 4.2 (4.17) | 8.3 (2.95)
  Pain Scale: Week 70 (n=3,14) | 2.8 (2.78) | 6.5 (2.17)
  Pain Scale: Week 73 (n=3,12) | 0.0 (0.00) | 9.7 (3.95)
  Pain Scale: Week 76 (n=3,8) | 5.6 (5.56) | 5.2 (2.19)
  Pain Scale: Week 79 (n=3,9) | 2.8 (2.78) | 7.4 (3.79)
  Pain Scale: Week 82 (n=2,6) | 0.0 (0.00) | 6.9 (3.98)
  Pain Scale: Week 85 (n=2,6) | 4.2 (4.17) | 5.6 (4.12)
  Pain Scale: Week 88 (n=2,6) | 8.3 (8.33) | 5.6 (2.78)
  Pain Scale: Week 91 (n=2,6) | 0.0 (0.00) | 2.1 (2.08)
  Pain Scale: Week 94 (n=2,6) | 0.0 (0.00) | 5.6 (3.51)
  Pain Scale: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (3.73)
  Pain Scale: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.3 (2.08)
  Pain Scale: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (3.40)
  Pain Scale: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.3 (3.99)
  Pain Scale: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 4.2 (2.41)
  Pain Scale: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 10.0 (4.86)
  Pain Scale: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 4.2 (2.41)
  Pain Scale: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (3.73)
  Pain Scale: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 10.0 (4.86)
  Pain Scale: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (3.73)
  Pain Scale: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Pain Scale: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 11.1 (7.35)
  Pain Scale: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 13.9 (7.35)
  Pain Scale: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 12.5 (4.17)
  Pain Scale: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 8.3 (8.33)
  Pain Scale: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 8.3 (0.00)
  Pain Scale: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Pain Scale: Final Visit (n=157,160) | 24.7 (1.60) | 26.8 (2.02)
  Reflux Symptoms Scale: BL (n=275,287) | 18.3 (1.29) | 16.9 (1.12)
  Reflux Symptoms Scale: Week 4 (n=234,250) | 14.8 (1.14) | 16.0 (1.09)
  Reflux Symptoms Scale: Week 7 (n=180,220) | 12.8 (1.26) | 15.4 (1.20)
  Reflux Symptoms Scale: Week 10 (n=176,203) | 12.6 (1.29) | 13.5 (1.18)
  Reflux Symptoms Scale: Week 13 (n=152,182) | 12.8 (1.39) | 12.9 (1.34)
  Reflux Symptoms Scale: Week 16 (n=120,165) | 12.0 (1.55) | 14.4 (1.58)
  Reflux Symptoms Scale: Week 19 (n=114,165) | 11.3 (1.76) | 10.6 (1.24)
  Reflux Symptoms Scale: Week 22 (n=79,143) | 9.0 (1.79) | 10.6 (1.37)
  Reflux Symptoms Scale: Week 25 (n=64,124) | 5.6 (1.21) | 9.7 (1.34)
  Reflux Symptoms Scale: Week 28 (n=47,111) | 6.6 (1.61) | 9.6 (1.42)
  Reflux Symptoms Scale: Week 31 (n=45,95) | 7.4 (1.69) | 10.1 (1.93)
  Reflux Symptoms Scale: Week 34 (n=45,95) | 7.2 (2.16) | 9.3 (1.77)
  Reflux Symptoms Scale: Week 37 (n=29,64) | 6.1 (1.62) | 10.9 (2.38)
  Reflux Symptoms Scale: Week 40 (n=24,55) | 7.9 (2.80) | 9.3 (2.13)
  Reflux Symptoms Scale: Week 43 (n=12,42) | 7.4 (3.44) | 9.0 (2.07)
  Reflux Symptoms Scale: Week 46 (n=14,42) | 4.8 (1.53) | 6.6 (1.97)
  Reflux Symptoms Scale: Week 49 (n=10,36) | 2.2 (1.48) | 6.5 (1.43)
  Reflux Symptoms Scale: Week 52 (n=8,30) | 2.8 (1.82) | 8.1 (2.55)
  Reflux Symptoms Scale: Week 55 (n=6,24) | 5.6 (5.56) | 6.5 (2.00)
  Reflux Symptoms Scale: Week 58 (n=6,21) | 0.0 (0.00) | 5.3 (1.65)
  Reflux Symptoms Scale: Week 61 (n=4,17) | 2.8 (2.78) | 2.6 (1.52)
  Reflux Symptoms Scale: Week 64 (n=3,20) | 3.7 (3.70) | 3.9 (1.85)
  Reflux Symptoms Scale: Week 67 (n=4,16) | 2.8 (2.78) | 6.3 (2.48)
  Reflux Symptoms Scale: Week 70 (n=3,13) | 3.7 (3.70) | 4.3 (2.00)
  Reflux Symptoms Scale: Week 73 (n=3,12) | 0.0 (0.00) | 7.9 (2.60)
  Reflux Symptoms Scale: Week 76 (n=3,8) | 3.7 (3.70) | 1.4 (1.39)
  Reflux Symptoms Scale: Week 79 (n=3,9) | 0.0 (0.00) | 3.7 (2.62)
  Reflux Symptoms Scale: Week 82 (n=2,6) | 0.0 (0.00) | 5.6 (2.48)
  Reflux Symptoms Scale: Week 85 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Reflux Symptoms Scale: Week 88 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Reflux Symptoms Scale: Week 91 (n=2,4) | 0.0 (0.00) | 0.0 (0.00)
  Reflux Symptoms Scale: Week 94 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Reflux Symptoms Scale: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 2.8 (2.78)
  Reflux Symptoms Scale: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 4.4 (4.44)
  Reflux Symptoms Scale: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (4.44)
  Reflux Symptoms Scale: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 7.4 (7.41)
  Reflux Symptoms Scale: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Reflux Symptoms Scale: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Reflux Symptoms Scale: Final Visit (n=1,5) | 15.3 (1.48) | 18.3 (1.72)
  Eating Restrictions (ER) Scale: BL (n=276,287) | 27.4 (1.44) | 23.9 (1.30)
  ER Scale: Week 4 (n=234,250) | 20.6 (1.24) | 21.1 (1.19)
  ER Scale: Week 7 (n=181,220) | 18.8 (1.36) | 19.0 (1.26)
  ER Scale: Week 10 (n=176,203) | 17.5 (1.25) | 17.4 (1.23)
  ER Scale: Week 13 (n=152,183) | 16.0 (1.77) | 17.0 (1.34)
  ER Scale: Week 16 (n=120,165) | 17.8 (1.77) | 15.1 (1.40)
  ER Scale: Week 19 (n=114,143) | 20.8 (2.01) | 15.5 (1.53)
  ER Scale: Week 22 (n=79,143) | 15.5 (2.14) | 13.6 (1.56)
  ER Scale: Week 25 (n=64,124) | 11.6 (2.14) | 12.9 (1.39)
  ER Scale: Week 28 (n=47,111) | 13.9 (2.64) | 11.3 (1.37)
  ER Scale: Week 31 (n=45,95) | 13.4 (2.69) | 12.5 (2.03)
  ER Scale: Week 34 (n=37,87) | 10.6 (2.16) | 10.9 (1.90)
  ER Scale: Week 37 (n=29,64) | 12.5 (3.10) | 9.5 (2.11)
  ER Scale: Week 40 (n=24,55) | 13.5 (3.32) | 9.5 (2.21)
  ER Scale: Week 43 (n=12,43) | 9.7 (3.22) | 7.0 (1.88)
  ER Scale: Week 46 (n=14,42) | 10.9 (3.07) | 6.0 (1.31)
  ER Scale: Week 49 (n=10,36) | 11.7 (3.09) | 8.1 (1.83)
  ER Scale: Week 52 (n=8,30) | 5.2 (2.19) | 9.3 (2.31)
  ER Scale: Week 55 (n=6,24) | 8.3 (4.30) | 5.2 (1.86)
  ER Scale: Week 58 (n=6,21) | 9.7 (5.45) | 6.0 (2.31)
  ER Scale: Week 61 (n=4,17) | 4.2 (2.41) | 5.4 (2.01)
  ER Scale: Week 64 (n=3,20) | 0.0 (0.00) | 8.3 (2.42)
  ER Scale: Week 67 (n=4,16) | 8.3 (4.81) | 10.4 (3.36)
  ER Scale: Week 70 (n=3,14) | 2.8 (2.78) | 6.5 (2.34)
  ER Scale: Week 73 (n=3,12) | 5.6 (5.56) | 9.0 (3.32)
  ER Scale: Week 76 (n=3,8) | 2.8 (2.78) | 5.2 (3.50)
  ER Scale: Week 79 (n=3,9) | 5.6 (5.56) | 5.6 (3.11)
  ER Scale: Week 82 (n=2,6) | 4.2 (4.17) | 2.8 (2.78)
  ER Scale: Week 85 (n=2,6) | 4.2 (4.17) | 4.2 (2.85)
  ER Scale: Week 88 (n=2,6) | 4.2 (4.17) | 4.2 (1.86)
  ER Scale: Week 91 (n=2,4) | 8.3 (8.33) | 4.2 (4.17)
  ER Scale: Week 94 (n=2,6) | 0.0 (0.00) | 4.2 (2.85)
  ER Scale: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (3.12)
  ER Scale: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.3 (3.99)
  ER Scale: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.3 (3.99)
  ER Scale: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 4.2 (4.17)
  ER Scale: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 4.2 (4.17)
  ER Scale: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 3.3 (3.33)
  ER Scale: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 4.2 (4.17)
  ER Scale: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (3.12)
  ER Scale: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 5.0 (3.33)
  ER Scale: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 1.7 (1.67)
  ER Scale: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  ER Scale: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 8.3 (4.81)
  ER Scale: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 5.6 (2.78)
  ER Scale: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  ER Scale: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 4.2 (4.17)
  ER Scale: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  ER Scale: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  ER Scale: Final Visit (n=157,160) | 23.8 (1.85) | 22.8 (1.84)
  Anxiety Scale: BL (n=276,287) | 47.5 (1.66) | 48.2 (1.54)
  Anxiety Scale: Week 4 (n=234,250) | 42.0 (1.66) | 43.8 (1.60)
  Anxiety Scale: Week 7 (n=181,220) | 40.6 (1.77) | 39.3 (1.66)
  Anxiety Scale: Week 10 (n=176,203) | 38.2 (1.98) | 38.2 (1.70)
  Anxiety Scale: Week 13 (n=152,183) | 35.7 (2.01) | 37.5 (1.99)
  Anxiety Scale: Week 16 (n=120,165) | 32.9 (2.27) | 37.1 (2.10)
  Anxiety Scale: Week 19 (n=114,143) | 35.8 (2.40) | 34.9 (2.04)
  Anxiety Scale: Week 22 (n=79,143) | 31.7 (3.16) | 32.8 (2.05)
  Anxiety Scale: Week 25 (n=64,124) | 25.2 (2.86) | 29.2 (2.03)
  Anxiety Scale: Week 28 (n=47,111) | 27.4 (3.65) | 26.9 (1.88)
  Anxiety Scale: Week 31 (n=45,95) | 29.1 (4.36) | 28.4 (2.32)
  Anxiety Scale: Week 34 (n=37,87) | 23.1 (3.69) | 27.8 (2.33)
  Anxiety Scale: Week 37 (n=29,64) | 27.2 (4.79) | 28.2 (2.87)
  Anxiety Scale: Week 40 (n=24,55) | 29.6 (3.99) | 26.3 (2.77)
  Anxiety Scale: Week 43 (n=12,43) | 30.6 (7.63) | 25.1 (2.91)
  Anxiety Scale: Week 46 (n=14,42) | 26.2 (6.34) | 23.3 (3.00)
  Anxiety Scale: Week 49 (n=14,42) | 20.0 (7.55) | 25.9 (3.03)
  Anxiety Scale: Week 52 (n=8,30) | 23.6 (7.98) | 27.4 (4.15)
  Anxiety Scale: Week 55 (n=6,24) | 31.5 (12.31) | 28.2 (3.90)
  Anxiety Scale: Week 58 (n=6,21) | 20.4 (10.11) | 21.7 (3.38)
  Anxiety Scale: Week 61 (n=4,17) | 8.3 (5.32) | 25.5 (5.37)
  Anxiety Scale: Week 64 (n=3,20) | 5.6 (5.56) | 23.9 (4.21)
  Anxiety Scale: Week 67 (n=4,16) | 11.1 (6.42) | 18.8 (3.47)
  Anxiety Scale: Week 70 (n=3,14) | 3.7 (3.70) | 27.0 (5.91)
  Anxiety Scale: Week 73 (n=3,12) | 7.4 (7.41) | 28.7 (6.03)
  Anxiety Scale: Week 76 (n=3,8) | 0.0 (0.00) | 27.8 (8.13)
  Anxiety Scale: Week 79 (n=3,9) | 11.1 (11.11) | 33.3 (8.28)
  Anxiety Scale: Week 82 (n=2,6) | 11.1 (11.11) | 25.9 (8.92)
  Anxiety Scale: Week 85 (n=2,6) | 11.1 (11.11) | 24.1 (3.41)
  Anxiety Scale: Week 88 (n=2,6) | 11.1 (11.11) | 14.8 (5.49)
  Anxiety Scale: Week 91 (n=2,4) | 11.1 (11.11) | 22.2 (4.54)
  Anxiety Scale: Week 94 (n=2,6) | 5.6 (5.56) | 22.2 (2.87)
  Anxiety Scale: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 31.1 (5.44)
  Anxiety Scale: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (5.56)
  Anxiety Scale: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 22.2 (4.54)
  Anxiety Scale: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 19.4 (5.32)
  Anxiety Scale: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (7.17)
  Anxiety Scale: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 22.2 (4.97)
  Anxiety Scale: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 19.4 (8.33)
  Anxiety Scale: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 20.0 (6.48)
  Anxiety Scale: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 15.6 (7.54)
  Anxiety Scale: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 17.8 (5.67)
  Anxiety Scale: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 22.2 (11.11)
  Anxiety Scale: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 18.5 (9.80)
  Anxiety Scale: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 18.5 (9.80)
  Anxiety Scale: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 16.7 (16.67)
  Anxiety Scale: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 11.1 (11.11)
  Anxiety Scale: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 16.7 (16.67)
  Anxiety Scale: Week 145 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Anxiety Scale: Final Visit (n=157,160) | 41.5 (2.19) | 40.9 (2.22)
  Dry Mouth: BL (n=274,287) | 24.5 (1.70) | 23.9 (1.70)
  Dry Mouth: Week 4 (n=232,249) | 24.0 (1.81) | 23.3 (1.59)
  Dry Mouth: Week 7 (n=180,219) | 24.6 (2.02) | 26.9 (1.87)
  Dry Mouth: Week 10 (n=176,203) | 23.5 (1.85) | 25.0 (1.96)
  Dry Mouth: Week 13 (n=152,183) | 23.2 (2.06) | 21.1 (1.95)
  Dry Mouth: Week 16 (n=120,165) | 23.9 (2.41) | 23.4 (2.19)
  Dry Mouth: Week 19 (n=113,143) | 22.4 (2.56) | 20.5 (2.17)
  Dry Mouth: Week 22 (n=79,143) | 19.0 (2.92) | 16.3 (2.06)
  Dry Mouth: Week 25 (n=64,124) | 16.1 (3.06) | 12.1 (1.80)
  Dry Mouth: Week 28 (n=47,111) | 10.6 (2.51) | 10.8 (1.55)
  Dry Mouth: Week 31 (n=45,95) | 12.6 (3.23) | 11.2 (2.21)
  Dry Mouth: Week 34 (n=37,87) | 9.9 (3.38) | 9.6 (1.88)
  Dry Mouth: Week 37 (n=29,64) | 12.6 (4.19) | 9.4 (2.28)
  Dry Mouth: Week 40 (n=23,55) | 8.7 (3.76) | 7.3 (2.40)
  Dry Mouth: Week 43 (n=12,43) | 11.1 (4.74) | 6.2 (2.00)
  Dry Mouth: Week 46 (n=14,42) | 9.5 (4.18) | 4.8 (1.82)
  Dry Mouth: Week 49 (n=10,36) | 16.7 (5.56) | 6.5 (2.23)
  Dry Mouth: Week 52 (n=8,30) | 12.5 (6.10) | 10.0 (3.26)
  Dry Mouth: Week 55 (n=6,24) | 5.6 (5.56) | 8.3 (3.01)
  Dry Mouth: Week 58 (n=6,21) | 11.1 (7.03) | 14.3 (4.35)
  Dry Mouth: Week 61 (n=4,17) | 8.3 (8.33) | 11.8 (4.90)
  Dry Mouth: Week 64 (n=3,20) | 0.0 (0.00) | 6.7 (3.06)
  Dry Mouth: Week 67 (n=4,16) | 8.3 (8.33) | 8.3 (4.81)
  Dry Mouth: Week 70 (n=3,14) | 0.0 (0.00) | 11.9 (5.64)
  Dry Mouth: Week 73 (n=3,12) | 0.0 (0.00) | 13.9 (4.95)
  Dry Mouth: Week 76 (n=3,8) | 0.0 (0.00) | 20.8 (8.77)
  Dry Mouth: Week 79 (n=3,9) | 0.0 (0.00) | 11.1 (5.56)
  Dry Mouth: Week 82 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Dry Mouth: Week 85 (n=2,6) | 16.7 (16.67) | 0.0 (0.00)
  Dry Mouth: Week 88 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Dry Mouth: Week 91 (n=2,4) | 0.0 (0.00) | 0.0 (0.00)
  Dry Mouth: Week 94 (n=2,6) | 0.0 (0.00) | 0.0 (0.00)
  Dry Mouth: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.0)
  Dry Mouth: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Dry Mouth: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Dry Mouth: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Dry Mouth: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Dry Mouth: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Dry Mouth: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Dry Mouth: Final Visit (n=157,157) | 24.0 (2.52) | 23.6 (2.43)
  Taste: BL (n=275,286) | 17.2 (1.56) | 17.9 (1.64)
  Taste: Week 4 (n=234,249) | 20.7 (1.63) | 24.8 (1.79)
  Taste: Week 7 (n=179,217) | 20.1 (1.78) | 24.0 (1.85)
  Taste: Week 10 (n=176,200) | 21.8 (1.86) | 25.3 (2.01)
  Taste: Week 13 (n=151,181) | 19.9 (2.08) | 25.2 (2.20)
  Taste: Week 16 (n=119,165) | 20.4 (2.22) | 23.8 (2.23)
  Taste: Week 19 (n=113,143) | 24.5 (2.37) | 22.6 (2.26)
  Taste: Week 22 (n=79,143) | 19.0 (2.86) | 19.6 (2.15)
  Taste: Week 25 (n=64,124) | 10.9 (2.23) | 15.9 (1.96)
  Taste: Week 28 (n=47,111) | 12.1 (2.76) | 14.7 (2.03)
  Taste: Week 31 (n=45,95) | 8.1 (2.63) | 13.0 (2.65)
  Taste: Week 34 (n=37,87) | 6.3 (2.53) | 9.6 (2.10)
  Taste: Week 37 (n=28,64) | 8.3 (3.26) | 7.8 (2.20)
  Taste: Week 40 (n=24,55) | 8.3 (3.01) | 7.9 (2.73)
  Taste: Week 43 (n=12,43) | 5.6 (3.75) | 7.0 (2.09)
  Taste: Week 46 (n=14,42) | 4.8 (3.24) | 7.9 (2.74)
  Taste: Week 49 (n=9,36) | 7.4 (4.90) | 4.6 (1.95)
  Taste: Week 52 (n=8,30) | 4.2 (4.17) | 7.8 (3.46)
  Taste: Week 55 (n=6,24) | 11.1 (7.03) | 4.2 (2.30)
  Taste: Week 58 (n=6,21) | 11.1 (7.03) | 4.8 (2.61)
  Taste: Week 61 (n=4,17) | 8.3 (8.33) | 0.0 (0.00)
  Taste: Week 64 (n=3,20) | 11.1 (11.11) | 1.7 (1.67)
  Taste: Week 67 (n=4,16) | 8.3 (8.33) | 4.2 (2.85)
  Taste: Week 70 (n=3,14) | 0.0 (0.00) | 0.0 (0.00)
  Taste: Week 73 (n=3,12) | 0.0 (0.00) | 2.8 (2.78)
  Taste: Week 76 (n=3,8) | 0.0 (0.00) | 0.0 (0.00)
  Taste: Week 79 (n=3,9) | 0.0 (0.00) | 0.0 (0.00)
  Taste: Week 82 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Taste: Week 85 (n=2, 6) | 0.0 (0.00) | 0.0 (0.00)
  Taste: Week 88 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Taste: Week 91 (n=2,4) | 0.0 (0.00) | 0.0 (0.00)
  Taste: Week 94 (n=2,6) | 0.0 (0.00) | 5.6 (5.56)
  Taste: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Taste: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Taste: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Taste: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Taste: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Taste: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Taste: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Taste: Final Visit (n=157,158) | 25.3 (2.26) | 20.3 (2.28)
  Body Image: BL (n=272,286) | 30.9 (1.95) | 31.9 (1.93)
  Body Image: Week 4 (n=233,249) | 32.6 (2.10) | 31.7 (2.03)
  Body Image: Week 7 (n=180,219) | 30.7 (2.19) | 27.9 (1.94)
  Body Image: Week 10 (n=175,203) | 30.1 (2.27) | 28.4 (2.05)
  Body Image: Week 13 (n=152,182) | 28.9 (2.54) | 28.2 (2.36)
  Body Image: Week 16 (n=119,165) | 29.1 (2.69) | 28.1 (2.29)
  Body Image: Week 19 (n=114,140) | 30.7 (2.82) | 25.0 (2.53)
  Body Image: Week 22 (n=79,143) | 28.7 (3.59) | 22.4 (2.29)
  Body Image: Week 25 (n=64,124) | 22.4 (3.32) | 22.6 (2.60)
  Body Image: Week 28 (n=47,111) | 23.4 (4.41) | 20.1 (2.53)
  Body Image: Week 31 (n=45,95) | 25.2 (4.87) | 19.3 (2.80)
  Body Image: Week 34 (n=37,87) | 18.9 (4.75) | 18.0 (2.66)
  Body Image: Week 37 (n=29,64) | 23.0 (5.99) | 18.2 (3.48)
  Body Image: Week 40 (n=24,55) | 20.8 (5.96) | 19.4 (3.53)
  Body Image: Week 43 (n=12,43) | 27.8 (6.91) | 15.5 (3.90)
  Body Image: Week 46 (n=14,42) | 21.4 (6.64) | 15.9 (3.81)
  Body Image: Week 49 (n=10,36) | 16.7 (7.45) | 13.9 (4.07)
  Body Image: Week 52 (n=8,30) | 16.7 (8.91) | 16.7 (3.83)
  Body Image: Week 55 (n=6,24) | 16.7 (11.39) | 16.7 (4.91)
  Body Image: Week 58 (n=6,21) | 11.1 (7.03) | 15.9 (5.45)
  Body Image: Week 61 (n=4,17) | 8.3 (8.33) | 13.7 (5.76)
  Body Image: Week 64 (n=3,20) | 0.0 (0.00) | 18.3 (4.51)
  Body Image: Week 67 (n=4,16) | 0.0 (0.00) | 14.6 (4.27)
  Body Image: Week 70 (n=4,14) | 0.0 (0.00) | 16.7 (5.79)
  Body Image: Week 73 (n=3,12) | 0.0 (0.00) | 27.8 (9.02)
  Body Image: Week 76 (n=3,8) | 0.0 (0.00) | 37.5 (11.68)
  Body Image: Week 79 (n=3,9) | 0.0 (0.00) | 25.9 (9.26)
  Body Image: Week 82 (n=2,6) | 0.0 (0.00) | 16.7 (7.45)
  Body Image: Week 85 (n=2,6) | 0.0 (0.00) | 11.1 (7.03)
  Body Image: Week 88 (n=2,5) | 0.0 (0.00) | 6.7 (6.67)
  Body Image: Week 91 (n=2,4) | 0.0 (0.00) | 16.7 (9.62)
  Body Image: Week 94 (n=2,6) | 0.0 (0.00) | 16.7 (7.45)
  Body Image: Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 13.3 (8.16)
  Body Image: Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Body Image: Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Body Image: Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (9.62)
  Body Image: Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 8.3 (8.33)
  Body Image: Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Body Image: Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (9.62)
  Body Image: Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Body Image: Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Body Image: Week 124 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.67 (6.67)
  Body Image: Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (11.11)
  Body Image: Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Body Image: Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 11.1 (11.11)
  Body Image: Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 16.7 (16.67)
  Body Image: Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Body Image: Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 16.7 (16.67)
  Body Image: Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Body Image: Final Visit (n=157,159) | 31.0 (2.58) | 30.4 (2.42)
  Hair Loss: BL (n=64,76) | 15.1 (3.31) | 25.0 (3.80)
  Hair Loss: Week 4 (n=68,71) | 20.1 (3.43) | 16.4 (2.90)
  Hair Loss: Week 7 (n=65,82) | 25.1 (3.27) | 19.1 (3.01)
  Hair Loss: Week 10 (n=75,78) | 21.8 (3.07) | 20.1 (2.81)
  Hair Loss: Week 13 (n=66,80) | 22.2 (3.40) | 20.4 (3.05)
  Hair Loss: Week 16 (n=53,72) | 28.3 (4.34) | 23.6 (3.26)
  Hair Loss: Week 19 (n=50,56) | 23.3 (4.29) | 21.4 (3.55)
  Hair Loss: Week 22 (n=38,54) | 20.2 (4.45) | 22.2 (3.52)
  Hair Loss: Week 25 (n=24,49) | 13.9 (4.88) | 18.4 (3.64)
  Hair Loss: Week 28 (n=20,39) | 26.7 (7.87) | 14.5 (4.38)
  Hair Loss: Week 31 (n=17,26) | 15.7 (7.07) | 10.3 (4.44)
  Hair Loss: Week 34 (n=13,24) | 7.7 (5.54) | 16.7 (5.68)
  Hair Loss: Week 37 (n=12,16) | 8.3 (5.98) | 12.5 (4.17)
  Hair Loss: Week 40 (n=11,13) | 12.1 (6.78) | 12.8 (6.01)
  Hair Loss: Week 43 (n=5,9) | 6.7 (6.67) | 3.7 (3.70)
  Hair Loss: Week 46 (n=5,13) | 26.7 (19.44) | 5.1 (3.47)
  Hair Loss: Week 49 (n=4,7) | 0.0 (0.00) | 9.5 (6.15)
  Hair Loss: Week 52 (n=3,4) | 11.1 (11.11) | 8.3 (8.33)
  Hair Loss: Week 55 (n=2,6) | 16.7 (16.67) | 0.0 (0.00)
  Hair Loss: Week 58 (n=2,3) | 16.7 (16.67) | 0.0 (0.00)
  Hair Loss: Week 61 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 16.7 (16.67)
  Hair Loss: Week 64 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 67 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 70 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 73 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.7 (6.67)
  Hair Loss: Week 76 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 79 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 82 (n=1,1) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Hair Loss: Week 85 (n=1,1) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Hair Loss: Week 88 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 91 (n=1,1) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Hair Loss: Week 94 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 97 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 100 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 103 (n=1,1) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Hair Loss: Week 106 (n=1,1) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Hair Loss: Week 109 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (0.00)
  Hair Loss: Week 112 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 115 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 118 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 121 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 124 (n=1,2) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (0.00)
  Hair Loss: Week 127 (n=1,1) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Hair Loss: Week 130 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Hair Loss: Week 133 (n=1,1) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Hair Loss: Final Visit (n=61,60) | 23.0 (3.62) | 19.4 (3.29)

13. Secondary Outcome: Pain Intensity Scores as Assessed By Visual Analog Scale (VAS)
Description: The participant assessed their pain on a 0 to 100 millimeter (mm) horizontal VAS. The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change indicated improvement.
Time Frame: as for outcome 11
Population: FAS; n = number of participants assessed for a specific parameter at a given visit.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
mm
  BL (n=275,284) | 21.1 (1.42) | 17.9 (1.25)
  Week 4 (n=234,249) | 14.6 (1.17) | 13.3 (1.11)
  Week 7 (n=181,219) | 11.1 (1.15) | 13.8 (1.31)
  Week 10 (n=174, 202) | 14.5 (1.46) | 12.9 (1.30)
  Week 13 (n=152,181) | 11.3 (1.37) | 12.2 (1.35)
  Week 16 (n=121,165) | 14.0 (1.77) | 12.8 (1.53)
  Week 19 (n=114,142) | 15.4 (1.92) | 12.0 (1.43)
  Week 22 (n=79,141) | 13.3 (2.20) | 15.1 (1.81)
  Week 25 (n=64,124) | 12.7 (2.39) | 11.0 (1.50)
  Week 28 (n=47,111) | 8.6 (1.85) | 12.3 (1.80)
  Week 31 (n=45,95) | 8.7 (2.11) | 12.5 (1.92)
  Week 34 (n=37,86) | 9.4 (2.90) | 10.7 (1.79)
  Week 37 (n=29,64) | 15.5 (4.08) | 10.9 (2.22)
  Week 40 (n=24,54) | 16.4 (4.20) | 8.8 (1.99)
  Week 43 (n=12,43) | 12.6 (5.04) | 7.2 (2.15)
  Week 46 (n=14,41) | 16.1 (6.11) | 7.4 (2.30)
  Week 49 (n=10,36) | 7.2 (3.71) | 6.5 (2.09)
  Week 52 (n=8,30) | 5.8 (3.43) | 6.9 (2.75)
  Week 55 (n=6,24) | 2.3 (1.20) | 3.3 (1.48)
  Week 58 (n=6,20) | 4.7 (2.20) | 3.8 (1.91)
  Week 61 (n=4,17) | 5.3 (3.04) | 7.2 (5.03)
  Week 64 (n=3,20) | 2.0 (1.00) | 6.8 (3.14)
  Week 67 (n=4,17) | 1.5 (0.96) | 8.9 (5.04)
  Week 70 (n=3,13) | 1.3 (1.33) | 1.3 (1.15)
  Week 73 (n=3,10) | 1.0 (0.58) | 16.5 (8.30)
  Week 76 (n=3,8) | 1.7 (0.88) | 12.9 (11.12)
  Week 79 (n=3,9) | 1.0 (0.58) | 5.9 (3.89)
  Week 82 (n=2,6) | 0.0 (0.00) | 4.8 (4.83)
  Week 85 (n=2,6) | 1.0 (1.00) | 6.3 (6.14)
  Week 88 (n=2,6) | 0.5 (0.50) | 5.7 (5.47)
  Week 91 (n=2,4) | 0.5 (0.50) | 7.5 (6.85)
  Week 94 (n=2,6) | 0.5 (0.50) | 5.8 (5.83)
  Week 97 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.2 (0.20)
  Week 100 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 0.3 (.25)
  Week 103 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.5 (5.85)
  Week 106 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 7.8 (6.79)
  Week 109 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 7.3 (7.25)
  Week 112 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 4.2 (3.50)
  Week 115 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 5.8 (5.11)
  Week 118 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 3.8 (3.32)
  Week 121 (n=1,5) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 3.2 (3.20)
  Week 124 (n=1,4) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 4.5 (3.84)
  Week 127 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 6.3 (6.33)
  Week 130 (n=0,3) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 5.7 (5.67)
  Week 133 (n=1,3) | 0.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated. | 5.0 (5.00)
  Week 136 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 6.0 (6.00)
  Week 139 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 8.0 (8.00)
  Week 142 (n=0,2) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 7.5 (7.50)
  Week 145 (n=0,1) | NA (NA) — No participants were analyzed in this treatment group for this timepoint. | 15.0 (NA) — Only 1 participant was analyzed in this treatment group at this timepoint, therefore standard error of the mean could not be calculated.
  Final visit/withdrawal (n=157,161) | 23.8 (1.99) | 21.9 (2.18)

14. Secondary Outcome: Percentage of Participants With a Change in Analgesic Medication During the Study
Description: Analgesic medications were recorded throughout the study until disease progression.
Time Frame: as for outcome 11
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
percentage of participants
  Taking any analgesic medication | 29.0 | 29.3
  Discontinued at least 1 medication | 5.9 | 1.7
  Decreased dose of at least 1 medication | 0.3 | 0.3
  No change in any medication | 5.5 | 7.1
  Increased dose or added at least 1 medication | 17.2 | 20.1

15. Secondary Outcome: Body Weight (Kilograms [kg]) at BL
Time Frame: BL
Population: FAS
Measure: Median (Full Range); unit: kg
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 290 | 294
kg | 60 [28 to 105] | 61 [35 to 110]

16. Secondary Outcome: Percentage of Participants With Change From Baseline in Body Weight by Percentage Change in Weight
Description: Change in body weight was categorized as an increase of greater than (>)5 percent (%), no change (plus or minus [±]5%), decrease of >5-10%, or a decrease of >10% from BL to the end of study. Time windows were applied in order to assign visits to weight measurements, and the lowest post-screening value recorded was used for the analysis. The percentage change in weight from screening was summarized over time.
Time Frame: as for outcome 11
Population: FAS. 273 and 283 participants were analyzed in the Fluoropyrimidine, Cisplatin and Trastuzumab, Fluoropyrimidine, Cisplatin groups, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 273 | 283
percentage of participants
  Increase >5% | 1.5 | 1.1
  No change (±5%) | 51.6 | 50.5
  Decrease >5-10% | 28.2 | 27.2
  Decrease >10% | 18.7 | 21.2

17. Secondary Outcome: Steady State Trastuzumab Area Under the Concentration (AUC)
Description: Individual steady state predicted exposure, as assessed by median AUC (measured as mg multiplied by [*] day per liter [L]) calculated for all treated participants using the nominal dosage schedule administered as an IV infusion. Individual steady state AUC was calculated using all available PK samples from all timepoints.
Time Frame: Predose and end of infusion on Days 1, 8, 15, and 64, and predose on Days 22 and 106
Population: Pharmacokinetic (PK) population: all participants with at least 1 measurement of trastuzumab serum concentration associated with a documented trastuzumab dosing history.
Measure: Median (90% Confidence Interval); unit: mg*day/L
Arm/Group | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 266
mg*day/L | 1030 [565 to 1726]

18. Secondary Outcome: Trastuzumab Minimum Serum Concentration (Cmin)
Description: Median Cmin (measured as milligrams per liter [mg/L]) calculated for all treated participants using the nominal dosage schedule administered as an IV infusion.
Time Frame: Predose and end of infusion on Days 1, 8, 15, and 64, and predose on Days 22 and 106
Population: PK Population
Measure: Median (90% Confidence Interval); unit: mg/L
Arm/Group | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 266
mg/L | 23.0 [6.4 to 48.5]

19. Secondary Outcome: Trastuzumab Maximum Serum Concentration (Cmax)
Description: Median Cmax (measured as mg/L) calculated for all treated participants using the nominal dosage schedule administered as an IV infusion.
Time Frame: Predose and end of infusion on Days 1, 8, 15, and 64, and predose on Days 22 and 106
Population: PK Population
Measure: Median (90% Confidence Interval); unit: mg/L
Arm/Group | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Number analyzed (Participants) | 266
mg/L | 128 [93.1 to 178]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from study start to 6 months after treatment completion. Drug-related Serious Adverse Events are collected through study and follow-up regardless of the time elapsed, or if the study has been closed.
Description: The safety analysis population included all patients who received at least one dose of trial treatment and had at least one safety follow-up.
Arm/Group | Fluoropyrimidine/Cisplatin (FP) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H)
Serious Adverse Events (participants affected / at risk) | 81/290 | 106/294
Other Adverse Events (participants affected / at risk) | 279/290 | 286/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluoropyrimidine/Cisplatin (FP) (N=290) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H) (N=294)
Diarrhoea (Gastrointestinal disorders) | 6 | 18
Vomiting (Gastrointestinal disorders) | 3 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 9
Nausea (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Gastrointestinal haemorrage (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastric perforation (Gastrointestinal disorders) | 0 | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Peritonitus (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
lleus paralytic (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 11
Anaemia (Blood and lymphatic system disorders) | 7 | 4
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 6
Septic shock (Infections and infestations) | 5 | 1
Respiratory tract infection (Infections and infestations) | 1 | 3
Infection (Infections and infestations) | 1 | 1
Biliary sepsis (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pneumococcal infection (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Asthenia (General disorders) | 3 | 3
Mucosal inflammation (General disorders) | 3 | 2
Pyrexia (General disorders) | 2 | 6
Death (General disorders) | 1 | 4
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Ill-defined disorder (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 7
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Cerebral infarcation (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 2
Cerebral disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 3
Renal failure (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Weight decreased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Device migration (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Arthritis infective (Infections and infestations) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluoropyrimidine/Cisplatin (FP) (N=290) | Trastuzumab + Fluoropyrimidine/Cisplatin (FP + H) (N=294)
Nausea (Gastrointestinal disorders) | 189 | 200
Vomiting (Gastrointestinal disorders) | 135 | 146
Diarrhoea (Gastrointestinal disorders) | 82 | 102
Constipation (Gastrointestinal disorders) | 95 | 76
Stomatitis (Gastrointestinal disorders) | 45 | 73
Abdominal pain (Gastrointestinal disorders) | 41 | 45
Abdominal pain upper (Gastrointestinal disorders) | 21 | 32
Dyspepsia (Gastrointestinal disorders) | 17 | 20
Dysphagia (Gastrointestinal disorders) | 11 | 17
Neutropenia (Blood and lymphatic system disorders) | 164 | 157
Anaemia (Blood and lymphatic system disorders) | 63 | 83
Thrombocytopenia (Blood and lymphatic system disorders) | 34 | 47
Fatigue (General disorders) | 86 | 106
Asthenia (General disorders) | 53 | 59
Pyrexia (General disorders) | 36 | 53
Mucosal inflammation (General disorders) | 15 | 39
Oedema (General disorders) | 26 | 25
Oedema peripheral (General disorders) | 13 | 18
Chills (General disorders) | 0 | 23
Decreased appetite (Metabolism and nutrition disorders) | 137 | 138
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 21
Dehydration (Metabolism and nutrition disorders) | 11 | 15
Palmer-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 66 | 78
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 36
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 17 | 19
Rash (Skin and subcutaneous tissue disorders) | 13 | 17
Dizziness (Nervous system disorders) | 29 | 31
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 28
Neuropathy peripheral (Nervous system disorders) | 25 | 26
Dysgeusia (Nervous system disorders) | 16 | 28
Headache (Nervous system disorders) | 20 | 15
Weight decreased (Investigations) | 40 | 68
Creatinine renal clearance decreased (Investigations) | 19 | 24
Weight increased (Investigations) | 15 | 21
Hiccups (Respiratory, thoracic and mediastinal disorders) | 29 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 15
Renal impairment (Renal and urinary disorders) | 38 | 46
Nephropathy toxic (Renal and urinary disorders) | 12 | 18
Nasopharyngitis (Infections and infestations) | 17 | 40
Insomnia (Psychiatric disorders) | 22 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.